CLINICAL TRIAL: NCT02198651
Title: A Phase 4 Trial Assessing the ImPact of Residual Inflammation Detected Via Imaging TEchniques, Drug Levels and Patient Characteristics on the Outcome of Dose TaperIng of Adalimumab in Clinical Remission Rheumatoid ArThritis (RA) Subjects (PREDICTRA)
Brief Title: A Phase 4 Trial Assessing the ImPact of Residual Inflammation Detected Via Imaging TEchniques, Drug Levels and Patient Characteristics on the Outcome of Dose TaperIng of Adalimumab in Clinical Remission Rheumatoid ArThritis (RA) Subjects
Acronym: PREDICTRA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M14-500; 2014-001114-26 (EudraCT Number)
Record Dates: First submitted 2014-07-22; First posted 2014-07-24 (Estimated); Results first posted 2019-06-25 (Actual); Last update posted 2019-06-25 (Actual); Status verified 2019-06

CONDITIONS: Rheumatoid Arthritis; Musculoskeletal and Connective Tissue Diseases
Keywords: Rheumatoid Arthritis; Adalimumab; Taper; Flare; Arthritis; Anti-rheumatic drugs; Remission; Magnetic Resonance Imaging; Ultrasound; Biomarker; Drug Level; Reduced dose
MeSH Terms: conditions — Arthritis, Rheumatoid; Connective Tissue Diseases; Arthritis | interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Adalimumab 40 mg eow (Experimental): 40 mg adalimumab administered subcutaneously every other week (eow) from Week 0 to Week 4 (Lead-in Period)
  Interventions: Biological: Adalimumab
- Adalimumab Tapering (Active Comparator): 40 mg adalimumab administered subcutaneously every three weeks from Week 4 to Week 40 (Double-blind Period)
  Interventions: Biological: Adalimumab
- Adalimumab Withdrawal Arm (Placebo Comparator): Placebo administered subcutaneously every three weeks from Week 4 to Week 40 (Double-blind Period)
  Interventions: Other: Placebo
- Adalimumab 40 mg eow Rescue Arm (Experimental): 40 mg adalimumab administered subcutaneously every other week from Flare Week 0 to Flare Week 16 (Open-label Rescue Period)
  Interventions: Biological: Adalimumab

INTERVENTIONS:
Biological: Adalimumab — Pre-filled syringe, administered by subcutaneous injection
  Other Names: ABT-D2E7; Humira
  Arms: Adalimumab 40 mg eow; Adalimumab 40 mg eow Rescue Arm; Adalimumab Tapering
Other: Placebo — Pre-filled syringe, administered by subcutaneous injection in the Double-blind period
  Arms: Adalimumab Withdrawal Arm

SUMMARY:
The primary objective of the study was to investigate the association between residual disease activity at Baseline as detected by Magnetic Resonance Imaging (MRI) and the occurrence of flares in participants with rheumatoid arthritis (RA) randomized to an adalimumab dose tapering regimen controlled by adalimumab withdrawal.

DETAILED DESCRIPTION:
This was a Phase 4, multicenter, randomized, double-blind, parallel-group study. The study included a Screening period of up to 28 days (unless extended with justification approved by study-designated physician), a 4-week Lead-In Period with open label (OL) 40 mg adalimumab administered subcutaneously (sc) every other week (eow), and a randomized 36-week double-blind period with 40 mg adalimumab sc every 3 weeks (q3wks; tapering arm) or placebo sc q3wks (withdrawal arm). Participants were randomized in a 5:1 ratio (tapering arm: withdrawal arm) after confirmation of meeting the disease activity score (DAS) criteria. Participants who experienced a protocol-defined flare at any time were to enter a rescue arm with OL 40 mg adalimumab administered sc eow for 16 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Participant had a diagnosis of rheumatoid arthritis (RA) as defined by the 1987 revised American College of Rheumatology (ACR) classification criteria and/or the ACR /European League Against Rheumatism (EULAR) 2010 classification criteria (any duration since diagnosis).
2. Participant must have met the following criteria:

   * Must have been treated with adalimumab 40 mg subcutaneously every other week (sc eow) for at least 12 months prior to Week 0 Visit
   * Must have been treated with concomitant methotrexate (MTX) at a stable dose (oral, sc or intramuscular (im) at any dose) for at least 12 weeks prior to Week 0 Visit or if not on MTX, must have been treated with other allowed conventional synthetic disease-modifying anti-rheumatic drugs (csDMARDs) at a stable dose for at least 12 weeks prior to Week 0 Visit or if not treated with csDMARDs must maintain this regimen for at least 12 weeks prior to Week 0 Visit.
3. Participant must be in sustained clinical remission based on the following:

   * At least one documented 4 or 3 (if Patient's Global Assessment ; PGA is not available) variables Disease Activity Score 28 Erythrocyte sedimentation rate (DAS28 ESR) or DAS28 C-reactive protein (CRP) < 2.6 (or calculated based on documented components of the DAS28) in the participant's chart 6 months or longer prior to the Screening Visit;
   * 4 variables DAS28 (ESR) assessed at Screening < 2.6, with all components including ESR assessed at Screening.
4. If participant was receiving concomitant allowed csDMARDs (in addition or not to MTX) the dose must have been stable for at least 12 weeks prior to the Week 0 Visit (e.g., chloroquine, hydroxychloroquine, sulfasalazine, gold formulations [including auranofin, gold sodium thiomalate, and aurothioglucose] and/or leflunomide).
5. If participant was receiving concomitant oral corticosteroids, prednisone or equivalent must have been < 10 mg/day and the dose must have been stable for at least 4 weeks prior to the Week 0 Visit.
6. If participant was receiving concomitant non-steroidal anti-inflammatory drugs (NSAIDs), tramadol or other equivalent opioids and/or non-opioid analgesics, the dose and/or therapeutic scheme must have been stable for at least 4 weeks prior to the Week 0 Visit.
7. Participant must have been able and willing to provide written informed consent and comply with the requirements of this study protocol.

Exclusion Criteria:

1. Any 4 or 3 (if PGA is not available) variables DAS28 (ESR) or DAS28 (CRP) (or calculated based on documented components of the DAS28) assessed within 6 months prior to the Screening Visit ≥ 2.6.
2. Participant was on an additional concomitant biological disease-modifying anti-rheumatic drug (bDMARD) (including but not limited to abatacept, anakinra, certolizumab, etanercept, golimumab, infliximab, rituximab or tocilizumab).
3. Participant had been treated with intra-articular or parenteral corticosteroids within the last four weeks before Screening.
4. Participant had undergone joint surgery within 12 weeks of Screening (at joints to be assessed by magnetic resonance imaging (MRI) and/or ultrasound).
5. Participant had a medical condition precluding an MRI (e.g. magnetic activated implanted devices - cardiac pace-maker, insulin pump, neuro stimulators, etc. and metallic devices or fragments or clips in the eye, brain or spinal canal and in the hand/wrist undergoing MRI)
6. Participant had a medical condition precluding a contrast MRI with gadolinium [e.g. nephrogenic systemic fibrosis, previous anaphylactic/anaphylactoid reaction to gadolinium containing contrast agent, pregnancy or breast feeding, severe renal insufficiency with an estimated Glomerular Filtration Rate (eGFR) below 30 mL/min/1.73m^2 at Screening, hepato-renal syndrome, severe chronic liver function impairment]
7. Participant had been treated with any investigational drug of chemical or biologic nature within a minimum of 30 days or five half-lives (whichever is longer) of the drug prior to the Screening Visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2015-01-05 (Actual); Primary Completion 2018-05-03 (Actual); Study Completion 2018-08-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (70):
- United States (13):
  - J Michael Grelier Research /ID# 149772, Tuscaloosa, Alabama
  - Westlake Medical Research (WMR) Clinical Trials /ID# 155386, Thousand Oaks, California
  - University of Florida /ID# 144851, Jacksonville, Florida
  - North Georgia Rheumatology Grp /ID# 155225, Lawrenceville, Georgia
  - The Arthritis & Diabetes Clinic, Inc. /ID# 149017, Monroe, Louisiana
  - Aa Mrc Llc /Id# 151933, Grand Blanc, Michigan
  - North Mississippi Med Clinics /ID# 149443, Tupelo, Mississippi
  - Montefiore Medical Center /ID# 155013, The Bronx, New York
  - Shanahan Rheuma & Immuno /ID# 148689, Raleigh, North Carolina
  - Altoona Ctr Clinical Res /ID# 148448, Duncansville, Pennsylvania
  - Low Country Rheumatology, PA /ID# 154198, Summerville, South Carolina
  - West Tennessee Research Inst /ID# 148391, Jackson, Tennessee
  - Arthritis Centers of Texas /ID# 152843, Dallas, Texas
- Australia (4):
  - Royal Prince Alfred Hospital /ID# 154649, Camperdown, New South Wales
  - Optimus Clinical Research Pty. /ID# 133881, Kogarah, New South Wales
  - John Hunter Hospital /ID# 133884, Newcastle, New South Wales
  - Rheumatology Research Unit /ID# 133883, Maroochydore, Queensland
- AKH Wien /ID# 133885, Vienna, Vienna, Austria
- Canada (5):
  - St. Joseph's Healthcare /ID# 149233, Hamilton, Ontario
  - The Arthritis Program Res Grp /ID# 129056, Newmarket, Ontario
  - Institut de Rhum. de Montreal /ID# 129055, Montreal, Quebec
  - Groupe de Recherche en Maladies Osseuses /ID# 129057, Sainte-Foy, Quebec
  - CIUSSS de l'Estrie - CHUS /ID# 144839, Sherbrooke, Quebec
- France (4):
  - CHU de la miletrie /ID# 133928, Poitiers, Poitou-Charentes
  - CHU Amiens Picardie /ID# 144846, Amiens, Somme
  - Hospital Louis Pasteur /ID# 134708, Chartres
  - CHU de Grenoble - Albet Michal /ID# 135953, Grenoble
- Germany (8):
  - Asklepios Klinik /ID# 129146, Bad Abbach
  - Charité Universitätsmedizin Campus Mitte /ID# 129142, Berlin
  - Immanuel-Krankenhaus /ID# 129143, Buch
  - Krankenhaus Porz am Rhein /ID# 129147, Cologne
  - Rheumaforschungszentrum II /ID# 148554, Hamburg
  - Klinikum der Univ Munich /ID# 129144, Munich
  - Rheumazentrum Ratingen /ID# 129148, Ratingen
  - Rheumatologische Praxis /ID# 151979, Rendsburg
- Greece (3):
  - University General Hospital "Attikon" /ID# 134709, Athens, Attica
  - General Hospital of Athens /ID# 129202, Athens
  - General UH of Heraklion /ID# 134712, Heraklion
- Hungary (3):
  - Budai Irgalmasrendi Korhaz /ID# 134714, Budapest
  - Orszagos Reumatologiai es Fizi /ID# 134710, Budapest
  - Debreceni Egyetem Klinikai Koz /ID# 134715, Debrecen
- St Vincent's University Hosp /ID# 129210, Dublin, Ireland
- Italy (5):
  - AP Romano Umberto I /ID# 132895, Rome, Lazio
  - A.O. Univ Consorziale Policlin /ID# 133932, Bari
  - Azienda Istituto Gaetano Pini /ID# 132964, Milan
  - Fondazione IRCCS Policlinico /ID# 133886, Pavia
  - A.O.U.I. di Verona Policlinico /ID# 132973, Verona
- Netherlands (4):
  - Jan van Breemen Instituut /ID# 133887, Amsterdam
  - Rijnstate Hospital /ID# 129206, Arnhem
  - Medisch Centrum Leeuwarden /ID# 133888, Leeuwarden
  - UMC Utrecht /ID# 132896, Utrecht
- Spain (9):
  - Hospital Parc de Salut del Mar /ID# 148670, Barcelona
  - Hosp Sant J. Despi-Moises Brog /ID# 135368, Barcelona
  - Hospital Universitario Basurto /ID# 135529, Bilbao
  - Hosp Clinico Virgen Arrixaca /ID# 137020, El Palmar
  - Hospital General Universitario Gregorio Maranon /ID# 133889, Madrid
  - Hospital Universitario La Paz /ID# 135369, Madrid
  - Hospital Univ De Mostoles /ID# 134489, Móstoles
  - Complejo Hosp Santiago /ID# 133890, Santiago de Compostela
  - Hosp General Univ de Valencia /ID# 134488, Valencia
- Sweden (3):
  - Akademiska Sjukhuset /ID# 148669, Uppsala, Uppsala County
  - Uppsala University Hospital /ID# 133891, Uppsala
  - Vastmanlands Sjukhus /ID# 133892, Västerås
- United Kingdom (7):
  - Whipps Cross Univ Hospital /ID# 133893, London, London, City of
  - Guy's and St Thomas' NHS Found /ID# 132965, London, London, City of
  - Mid Essex Hospitals NHS Trust /ID# 151636, Chelmsford
  - Western General Hospital /ID# 132966, Edinburgh
  - Chapel Allerton Hospital /ID# 129208, Leeds
  - University Hospital Aintree /ID# 132980, Liverpool
  - Queen Alexandra Hospital /ID# 132982, Portsmouth

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- [Derived] Emery P, Burmester GR, Naredo E, Sinigaglia L, Lagunes I, Koenigsbauer F, Conaghan PG. Adalimumab dose tapering in patients with rheumatoid arthritis who are in long-standing clinical remission: results of the phase IV PREDICTRA study. Ann Rheum Dis. 2020 Aug;79(8):1023-1030. doi: 10.1136/annrheumdis-2020-217246. Epub 2020 May 13. PMID 32404343
- [Derived] Emery P, Burmester GR, Naredo E, Zhou Y, Hojnik M, Conaghan PG. Design of a phase IV randomised, double-blind, placebo-controlled trial assessing the ImPact of Residual Inflammation Detected via Imaging TEchniques, Drug Levels and Patient Characteristics on the Outcome of Dose TaperIng of Adalimumab in Clinical Remission Rheumatoid ArThritis (RA) patients (PREDICTRA). BMJ Open. 2018 Feb 28;8(2):e019007. doi: 10.1136/bmjopen-2017-019007. PMID 29490959
- See also: Related Info — https://www.rxabbvie.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All Lead-in-Treated Subject population: participants who were enrolled in the study and received at least 1 dose of study drug during the Lead-in period. Three participants enrolled in the study but were not treated during the Lead-in period.
Groups:
- Adalimumab Tapering to Rescue Arm; Adalimumab Withdrawal to Rescue Arm: 40 mg adalimumab administered subcutaneously every other week (eow) from Flare Week 0 to Flare Week 16 (Open-Label Rescue Period)
Period: Lead-in Period
Arm/Group | Adalimumab 40 mg Eow | Adalimumab Tapering | Adalimumab Withdrawal Arm | Adalimumab Tapering to Rescue Arm | Adalimumab Withdrawal to Rescue Arm
Started | 149 | 0 | 0 | 0 | 0
Participants Treated in Lead-In Period | 146 | 0 | 0 | 0 | 0
Completed | 112 | 0 | 0 | 0 | 0
Not Completed | 37 | 0 | 0 | 0 | 0
Not completed — Withdrew consent | 13 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 2 | 0 | 0 | 0 | 0
Not completed — Other, not specified | 22 | 0 | 0 | 0 | 0
Period: Double-blind Period
Arm/Group | Adalimumab 40 mg Eow | Adalimumab Tapering | Adalimumab Withdrawal Arm | Adalimumab Tapering to Rescue Arm | Adalimumab Withdrawal to Rescue Arm
Started | 0 | 102 | 20 | 0 | 0
Completed | 0 | 93 | 19 | 0 | 0
Not Completed | 0 | 9 | 1 | 0 | 0
Not completed — Withdrew consent | 0 | 4 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0
Not completed — Other, not specified | 0 | 4 | 1 | 0 | 0
Period: Open-label Rescue Period
Arm/Group | Adalimumab 40 mg Eow | Adalimumab Tapering | Adalimumab Withdrawal Arm | Adalimumab Tapering to Rescue Arm | Adalimumab Withdrawal to Rescue Arm
Started | 0 | 0 | 0 | 31 | 8
Correctly Entered Open-label Rescue | 0 | 0 | 0 | 30 | 8
Completed | 0 | 0 | 0 | 28 | 8
Not Completed | 0 | 0 | 0 | 3 | 0
Not completed — Withdrew consent | 0 | 0 | 0 | 2 | 0
Not completed — Incorrectly entered Open-label Rescue | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All Lead-in-Treated Subject population: participants who were enrolled in the study and received at least 1 dose of study drug during the Lead-in period
Arm/Group | Adalimumab 40 mg Eow
Number analyzed (Participants) | 146
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (10.30)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 109
  Male | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 139
  More than one race | 0
  Unknown or Not Reported | 3
Tobacco Use [Count of Participants; unit: Participants]
  Current | 22
  Former | 46
  Never | 76
  Unknown | 2
Disease duration [Mean (Standard Deviation); unit: years] — Population: Participants with available data
  years
    number analyzed (Participants) | 142
    (all) | 12.9 (9.99)
Duration of adalimumab therapy [Mean (Standard Deviation); unit: years] | 5.4 (3.27)
Duration of remission [Mean (Standard Deviation); unit: years] — Population: Participants with available data
  years
    number analyzed (Participants) | 125
    (all) | 2.2 (1.99)
Previous treatment with conventional synthetic disease-modifying anti-rheumatic drugs (csDMARDs) [Count of Participants; unit: Participants]
  Yes | 145
  No | 1
Previous Tx with biological disease-modifying anti-rheumatic drugs (bDMARDs; excluding adalimumab) [Count of Participants; unit: Participants]
  Yes | 38
  No | 108
Previous Tx with csDMARDS or bDMARDs (excluding adalimumab) [Count of Participants; unit: Participants]
  Yes | 146
  No | 0
Participants' Global Assessment of Disease Activity [Mean (Standard Deviation); unit: units on a scale] — Participants rated the severity of their rheumatoid arthritis symptoms and how well they were doing during the last 24 hours by placing a vertical mark on a line with a range of 0 (very well) to 100 mm (very poorly).
  units on a scale | 8.7 (11.84)
Mean C-Reactive Protein (CRP) [Mean (Standard Deviation); unit: mg/L] — C-Reactive Protein (CRP; mg/L) was measured from blood samples as a marker for inflammation.
  mg/L | 2.4 (2.58)
HAQ-DI Score [Mean (Standard Deviation); unit: units on a scale] — The Health Assessment Questionnaire- Disability Index (HAQ-DI) is specific for rheumatoid arthritis. 20 questions refer to eight domains:dressing/grooming, arising, eating, walking, hygiene, reach, grip, and daily activities. Participants rated their ability to do each task over the past 7 days: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task were summed and averaged to provide an overall score ranging from 0 to 3, where zero represents no disability and three very severe, high-dependency disability.
  units on a scale | 0.4 (0.51)

OUTCOME MEASURES:

1. Primary Outcome: Association Between Baseline Hand and Wrist Synovitis Rheumatoid Arthritis Magnetic Resonance Imaging Scoring System (RAMRIS) Score and Flare up to Week 40 in the Tapering Arm
Description: Synovitis was assessed in three wrist regions (the distal radioulnar joint; the radiocarpal joint; the intercarpal and carpometacarpal joints) and in each Metacarpophalangeal joint (MCP) joint. The first carpometacarpal joint and the first MCP joint are not scored. The scale is 0-3. Score 0 is normal, and 1-3 (mild, moderate, severe) are by thirds of the presumed maximum volume of enhancing tissue in the synovial compartment. Flare is defined as an increase from Double-blind Baseline in DAS (Disease Activity Score) 28 erythrocyte sedimentation rate (ESR) of > 0.6 AND DAS28 [ESR] > 2.6, OR an increase in DAS28 (ESR) of ≥ 1.2 irrespective of the resulting DAS28 [ESR]. The association between baseline hand and wrist synovitis RAMRIS score and occurrence of rheumatoid arthritis flare up to Week 40 in the Tapering arm was examined using logistic regression, and the 95% confidence interval of the odds ratio was calculated.
Time Frame: From Week 4 to Week 40
Population: Participants in the Tapering arm who received at least 1 dose of study drug during the Double-blind period
Measure: Number (95% Confidence Interval); unit: odds ratio
Arm/Group | Adalimumab Tapering
Number analyzed (Participants) | 102
odds ratio | 0.993 [0.822 to 1.199]
Statistical Analysis 1: Comparison: Adalimumab Tapering; Test type: Other; p = 0.943, Wald Chi

2. Primary Outcome: Association Between Baseline Bone Marrow Edema RAMRIS Score and Flare up to Week 40 in the Tapering Arm
Description: Bone marrow edema in each bone was scored separately. The scale is 0-3 based on the proportion of bone with edema, as follows-0: no edema; 1: 1-33% of bone edematous; 2: 34-66% of bone edematous; 3: 67-100%. Flare is defined as an increase from Double-blind Baseline in DAS (Disease Activity Score) 28 erythrocyte sedimentation rate (ESR) of > 0.6 AND DAS28 [ESR] > 2.6, OR an increase in DAS28 (ESR) of ≥ 1.2 irrespective of the resulting DAS28 [ESR]. The association between baseline bone marrow edema rheumatoid arthritis MRI scoring system (RAMRIS) score and occurrence of rheumatoid arthritis flare up to Week 40 in the Tapering arm was examined using logistic regression, and the 95% confidence interval of the odds ratio was calculated.
Time Frame: From Week 4 to Week 40
Population: Participants in the Tapering arm who received at least 1 dose of study drug during the Double-blind period
Measure: Number (95% Confidence Interval); unit: odds ratio
Arm/Group | Adalimumab Tapering
Number analyzed (Participants) | 102
odds ratio | 0.959 [0.821 to 1.119]
Statistical Analysis 1: Comparison: Adalimumab Tapering; Test type: Other; p = 0.592, Wald Chi

3. Primary Outcome: Association Between a Composite of Baseline Hand and Wrist Synovitis and Bone Marrow Edema RAMRIS Scores and Flare up to Week 40 in the Tapering Arm
Description: The composite score is the sum of the baseline hand and wrist synovitis and bone marrow edema RAMRIS scores. Flare is defined as an increase from Double-blind Baseline in DAS (Disease Activity Score) 28 erythrocyte sedimentation rate (ESR) of > 0.6 AND DAS28 [ESR] > 2.6, OR an increase in DAS28 (ESR) of ≥ 1.2 irrespective of the resulting DAS28 [ESR]. The association between the composite baseline hand and wrist synovitis score and baseline bone marrow edema rheumatoid arthritis MRI scoring system (RAMRIS) score and occurrence of rheumatoid arthritis flare up to Week 40 in the Tapering arm was examined using logistic regression, and the 95% confidence interval of the odds ratio was calculated.
Time Frame: From Week 4 to Week 40
Population: Participants in the Tapering arm who received at least 1 dose of study drug during the Double-blind period
Measure: Number (95% Confidence Interval); unit: odds ratio
Arm/Group | Adalimumab Tapering
Number analyzed (Participants) | 102
odds ratio | 0.979 [0.885 to 1.084]
Statistical Analysis 1: Comparison: Adalimumab Tapering; Test type: Other; p = 0.688, Wald Chi

4. Secondary Outcome: Median Time to Flare
Description: Time to flare was defined as the number of weeks from the date of the first dose of study drug in the Double-blind period to the date of flare.
Time Frame: From Week 4 to Week 40
Population: Double-blind Treated Subject population: participants who received at least 1 dose of study drug during the Double-blind period
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Adalimumab Tapering | Adalimumab Withdrawal Arm
Number analyzed (Participants) | 102 | 20
weeks | NA [36.4 to NA] — NA = not estimable/calculable due to low number of events | NA [12.1 to NA] — NA = not estimable/calculable due to low number of events

5. Secondary Outcome: Physicians' Assessment of Flare Severity
Description: Physicians rated the severity of flare at the Flare Week 0 visit from 0 (not severe) to 10 (very severe). The number of participants within each level of flare severity is presented.
Time Frame: At the Flare Week 0 Visit
Population: All Open-label-rescue-treated participants excluding those who falsely entered the Open-label rescue period
Measure: Count of Participants; unit: Participants
Arm/Group | Adalimumab Tapering | Adalimumab Withdrawal Arm
Number analyzed (Participants) | 30 | 8
Participants
  0 | 1 | 1
  1 | 2 | 0
  2 | 3 | 0
  3 | 3 | 1
  4 | 6 | 2
  5 | 1 | 1
  6 | 4 | 0
  7 | 1 | 0
  8 | 0 | 0
  9 | 0 | 0
  10 | 0 | 0
  Missing | 9 | 3

6. Secondary Outcome: Participants' Assessment of Flare Severity
Description: Participants rated the severity of flare at the Flare Week 0 visit from 0 (not severe) to 10 (very severe). The number of participants within each level of flare severity is presented.
Time Frame: At the Flare Week 0 Visit
Population: All Open-label-rescue-treated participants excluding those who falsely entered the Open-label rescue period
Measure: Count of Participants; unit: Participants
Arm/Group | Adalimumab Tapering | Adalimumab Withdrawal Arm
Number analyzed (Participants) | 30 | 8
Participants
  0 | 1 | 0
  1 | 2 | 1
  2 | 2 | 2
  3 | 3 | 0
  4 | 4 | 0
  5 | 1 | 1
  6 | 4 | 1
  7 | 1 | 0
  8 | 2 | 0
  9 | 0 | 0
  10 | 2 | 0
  Missing | 8 | 3

7. Secondary Outcome: Percentage of Participants With a Flare
Description: Flare was defined as an increase from Double-blind Baseline in DAS (Disease Activity Score) 28 erythrocyte sedimentation rate (ESR) of > 0.6 AND DAS28 [ESR] > 2.6, OR an increase in DAS28 (ESR) of ≥ 1.2 irrespective of the resulting DAS28 [ESR].
Time Frame: From Week 4 to Week 40
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Adalimumab Tapering | Adalimumab Withdrawal Arm
Number analyzed (Participants) | 102 | 20
percentage of participants | 36.3 [27.0 to 46.4] | 45.0 [23.1 to 68.5]

8. Secondary Outcome: Number of Participants Who Regained Clinical Remission in the Open-Label Rescue Arm Over Time
Description: The Disease Activity Score 28 (DAS28) is a validated index of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, the erythrocyte sedimentation rate (ESR; mm/hour), and the participant's assessment of global disease activity (on a visual analog scale [VAS] from 0 to 10 cm) are included in the DAS28 (ESR) score. Scores on the DAS28 range from 0 to 10; higher scores indicate more disease activity. Clinical remission was defined as DAS28 (ESR) < 2.6.
Time Frame: From Flare Week 0 to Flare Week 16
Population: All Open-label rescue-treated participants excluding those who incorrectly entered the Open-label Rescue Period; last observation carried forward
Measure: Count of Participants; unit: Participants
Arm/Group | Adalimumab Tapering | Adalimumab Withdrawal Arm
Number analyzed (Participants) | 30 | 8
Participants
  Flare Week 0 | 3 | 1
  Flare Week 4: number analyzed (Participants) | 29 | 7
  Flare Week 4 | 14 | 1
  Flare Week 10: number analyzed (Participants) | 29 | 7
  Flare Week 10 | 17 | 3
  Flare Week 16: number analyzed (Participants) | 29 | 8
  Flare Week 16 | 13 | 4

9. Secondary Outcome: Median Time to Clinical Remission From the Occurrence of Flare
Description: The Disease Activity Score 28 (DAS28) is a validated index of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, the erythrocyte sedimentation rate (ESR; mm/hour), and the participant's assessment of global disease activity (on a visual analog scale [VAS] from 0 to 10 cm) are included in the DAS28 (ESR) score. Scores on the DAS28 range from 0 to 10; higher scores indicate more disease activity. Clinical remission was defined as DAS28 (ESR) < 2.6. Time to clinical remission was defined as the number of weeks from the occurrence of flare to the first date of clinical remission.
Time Frame: From Flare Week 0 to Flare Week 16
Population: All Open-label rescue treated participants excluding those who incorrectly entered the Open-label Rescue Period
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Adalimumab Tapering | Adalimumab Withdrawal Arm
Number analyzed (Participants) | 30 | 8
weeks | 6.1 [4.1 to 16.3] | 18.0 [0.1 to 18.0]

10. Secondary Outcome: Mean Change From Double-blind Baseline in Disease Activity Score 28 (DAS28)
Description: The Disease Activity Score 28 (DAS28) is a validated index of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, the erythrocyte sedimentation rate (ESR; mm/hour), and the participant's assessment of global disease activity (on a visual analog scale [VAS] from 0 to 10 cm) are included in the DAS28 (ESR) score. Scores on the DAS28 range from 0 to 10; higher scores indicate more disease activity. Negative values indicate improvement from baseline.
Time Frame: From Week 4 to Week 40 and from Flare Week 0 to Flare Week 16
Population: Double-blind Treated Subject population: participants who received at least 1 dose of study drug during the Double-blind period and had at least Double-blind Baseline data for this endpoint
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Flared Participants: Participants who experienced flare during the Double-blind Period
- Non-Flared Participants: Participants who did not experience flare during the Double-blind Period
Arm/Group | Flared Participants | Non-Flared Participants
Number analyzed (Participants) | 46 | 76
units on a scale
  Double Blind Week 10- Tapering Arm: number analyzed (Participants) | 37 | 63
  Double Blind Week 10- Tapering Arm | 0.7 (1.27) | 0.1 (0.46)
  Double Blind Week 10- Withdrawal Arm: number analyzed (Participants) | 9 | 11
  Double Blind Week 10- Withdrawal Arm | 0.1 (0.47) | 0.1 (0.55)
  Double Blind Week 16- Tapering Arm: number analyzed (Participants) | 35 | 63
  Double Blind Week 16- Tapering Arm | 1.2 (1.34) | 0.1 (0.39)
  Double Blind Week 16- Withdrawal Arm: number analyzed (Participants) | 9 | 11
  Double Blind Week 16- Withdrawal Arm | 0.9 (0.58) | 0.0 (0.43)
  Double Blind Week 22- Tapering Arm: number analyzed (Participants) | 19 | 63
  Double Blind Week 22- Tapering Arm | 0.7 (1.18) | -0.0 (0.53)
  Double Blind Week 22- Withdrawal Arm: number analyzed (Participants) | 4 | 11
  Double Blind Week 22- Withdrawal Arm | 0.5 (0.31) | 0.1 (0.24)
  Double Blind Week 28- Tapering arm: number analyzed (Participants) | 16 | 63
  Double Blind Week 28- Tapering arm | 0.8 (1.16) | 0.1 (0.50)
  Double Blind Week 28- Withdrawal arm: number analyzed (Participants) | 4 | 11
  Double Blind Week 28- Withdrawal arm | 1.0 (1.54) | 0.2 (0.25)
  Double Blind Week 34- Tapering Arm: number analyzed (Participants) | 12 | 63
  Double Blind Week 34- Tapering Arm | 0.7 (0.59) | -0.0 (0.54)
  Double Blind Week 34- Withdrawal Arm: number analyzed (Participants) | 2 | 11
  Double Blind Week 34- Withdrawal Arm | -0.7 (0.11) | -0.0 (0.46)
  Double Blind Week 40- Tapering Arm: number analyzed (Participants) | 11 | 63
  Double Blind Week 40- Tapering Arm | 1.5 (1.20) | 0.0 (0.52)
  Double Blind Week 40- Withdrawal Arm: number analyzed (Participants) | 2 | 11
  Double Blind Week 40- Withdrawal Arm | 0.8 (2.18) | 0.2 (0.38)
  Flare Week 0- Tapering Arm: number analyzed (Participants) | 30 | 0
  Flare Week 0- Tapering Arm | 2.3 (1.15) |
  Flare Week 0- Withdrawal Arm: number analyzed (Participants) | 8 | 0
  Flare Week 0- Withdrawal Arm | 1.9 (0.96) |
  Flare Week 4- Tapering Arm: number analyzed (Participants) | 29 | 0
  Flare Week 4- Tapering Arm | 1.3 (1.05) |
  Flare Week 4- Withdrawal Arm: number analyzed (Participants) | 7 | 0
  Flare Week 4- Withdrawal Arm | 1.2 (1.14) |
  Flare Week 10- Tapering Arm: number analyzed (Participants) | 29 | 0
  Flare Week 10- Tapering Arm | 0.9 (0.81) |
  Flare Week 10- Withdrawal Arm: number analyzed (Participants) | 7 | 0
  Flare Week 10- Withdrawal Arm | 0.7 (0.50) |
  Flare Week 16- Tapering Arm: number analyzed (Participants) | 29 | 0
  Flare Week 16- Tapering Arm | 1.2 (1.04) |
  Flare Week 16- Withdrawal Arm: number analyzed (Participants) | 8 | 0
  Flare Week 16- Withdrawal Arm | 0.6 (0.80) |

11. Secondary Outcome: Mean Change From Double-blind Baseline in Clinical Disease Activity Index (CDAI) Score
Description: The CDAI is a validated measure of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, global health assessed by the participant on a visual analogue scale from 0 to 10 (cm), and global health assessed by an investigator on a visual analogue scale from 0 to 10 (cm) were included in the CDAI score. Scores on the CDAI range from 0 to 76; higher scores indicate more disease activity. Negative values indicate improvement from the Double-blind baseline score.
Time Frame: From Week 4 to Week 40 and from Flare Week 0 to Flare Week 16
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Flared Participants | Non-Flared Participants
Number analyzed (Participants) | 46 | 76
units on a scale
  Double Blind Week 10- Tapering Arm: number analyzed (Participants) | 37 | 62
  Double Blind Week 10- Tapering Arm | 4.4 (7.68) | 0.6 (1.34)
  Double Blind Week 10- Withdrawal Arm: number analyzed (Participants) | 9 | 11
  Double Blind Week 10- Withdrawal Arm | 1.0 (2.45) | 1.4 (2.85)
  Double Blind Week 16- Tapering Arm: number analyzed (Participants) | 35 | 63
  Double Blind Week 16- Tapering Arm | 7.0 (9.35) | 0.4 (1.30)
  Double Blind Week 16- Withdrawal Arm: number analyzed (Participants) | 9 | 11
  Double Blind Week 16- Withdrawal Arm | 2.9 (2.42) | -0.1 (0.88)
  Double Blind Week 22- Tapering Arm: number analyzed (Participants) | 19 | 63
  Double Blind Week 22- Tapering Arm | 3.2 (4.98) | 0.3 (1.38)
  Double Blind Week 22- Withdrawal Arm: number analyzed (Participants) | 4 | 11
  Double Blind Week 22- Withdrawal Arm | 2.2 (1.93) | 0.1 (0.73)
  Double Blind Week 28- Tapering arm: number analyzed (Participants) | 16 | 63
  Double Blind Week 28- Tapering arm | 3.7 (6.19) | 0.5 (1.37)
  Double Blind Week 28- Withdrawal arm: number analyzed (Participants) | 4 | 11
  Double Blind Week 28- Withdrawal arm | 6.3 (8.40) | -0.1 (0.80)
  Double Blind Week 34- Tapering Arm: number analyzed (Participants) | 12 | 63
  Double Blind Week 34- Tapering Arm | 2.7 (3.04) | 0.2 (1.08)
  Double Blind Week 34- Withdrawal Arm: number analyzed (Participants) | 2 | 11
  Double Blind Week 34- Withdrawal Arm | -0.1 (0.14) | 0.0 (0.92)
  Double Blind Week 40- Tapering Arm: number analyzed (Participants) | 11 | 63
  Double Blind Week 40- Tapering Arm | 7.4 (10.04) | 0.1 (1.33)
  Double Blind Week 40- Withdrawal Arm: number analyzed (Participants) | 2 | 11
  Double Blind Week 40- Withdrawal Arm | 7.7 (11.38) | -0.3 (0.48)
  Flare Week 0- Tapering Arm: number analyzed (Participants) | 30 | 0
  Flare Week 0- Tapering Arm | 12.3 (9.56) |
  Flare Week 0- Withdrawal Arm: number analyzed (Participants) | 8 | 0
  Flare Week 0- Withdrawal Arm | 9.4 (9.13) |
  Flare Week 4- Tapering Arm: number analyzed (Participants) | 28 | 0
  Flare Week 4- Tapering Arm | 5.0 (6.55) |
  Flare Week 4- Withdrawal Arm: number analyzed (Participants) | 7 | 0
  Flare Week 4- Withdrawal Arm | 5.4 (9.59) |
  Flare Week 10- Tapering Arm: number analyzed (Participants) | 29 | 0
  Flare Week 10- Tapering Arm | 3.5 (4.55) |
  Flare Week 10- Withdrawal Arm: number analyzed (Participants) | 7 | 0
  Flare Week 10- Withdrawal Arm | 3.6 (2.52) |
  Flare Week 16- Tapering Arm: number analyzed (Participants) | 29 | 0
  Flare Week 16- Tapering Arm | 4.5 (6.14) |
  Flare Week 16- Withdrawal Arm: number analyzed (Participants) | 8 | 0
  Flare Week 16- Withdrawal Arm | 2.8 (4.19) |

12. Secondary Outcome: Mean Change From Double-blind Baseline in Simplified Disease Activity Index (SDAI) Score
Description: The SDAI is a validated measure of rheumatoid arthritis disease activity. Twenty-eight tender joint counts, 28 swollen joint counts, global health assessed by the participant on a visual analogue scale from 0 to 10 (cm), global health assessed by an investigator on a visual analogue scale from 0 to 10 (cm), and serum levels of C-reactive protein levels (mg/dL) were included in the SDAI score. Scores on the SDAI range from 0 to 86; higher scores indicate more disease activity. Negative values indicate improvement from the Double-blind baseline score.
Time Frame: From Week 4 to Week 40 and from Flare Week 0 to Flare Week 16
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Flared Participants | Non-Flared Participants
Number analyzed (Participants) | 46 | 76
units on a scale
  Double Blind Week 10- Tapering Arm: number analyzed (Participants) | 36 | 62
  Double Blind Week 10- Tapering Arm | 3.7 (8.57) | 0.8 (1.85)
  Double Blind Week 10- Withdrawal Arm: number analyzed (Participants) | 9 | 11
  Double Blind Week 10- Withdrawal Arm | 0.9 (2.59) | 1.3 (2.67)
  Double Blind Week 16- Tapering Arm: number analyzed (Participants) | 35 | 63
  Double Blind Week 16- Tapering Arm | 6.3 (10.25) | 0.4 (1.35)
  Double Blind Week 16- Withdrawal Arm: number analyzed (Participants) | 9 | 11
  Double Blind Week 16- Withdrawal Arm | 3.6 (2.80) | -0.1 (0.90)
  Double Blind Week 22- Tapering Arm: number analyzed (Participants) | 19 | 63
  Double Blind Week 22- Tapering Arm | 3.6 (5.18) | 0.3 (1.47)
  Double Blind Week 22- Withdrawal Arm: number analyzed (Participants) | 4 | 11
  Double Blind Week 22- Withdrawal Arm | 2.3 (1.95) | -0.0 (0.88)
  Double Blind Week 28- Tapering arm: number analyzed (Participants) | 16 | 63
  Double Blind Week 28- Tapering arm | 3.8 (6.34) | 0.4 (1.37)
  Double Blind Week 28- Withdrawal arm: number analyzed (Participants) | 4 | 11
  Double Blind Week 28- Withdrawal arm | 6.4 (8.40) | 0.1 (1.61)
  Double Blind Week 34- Tapering Arm: number analyzed (Participants) | 12 | 63
  Double Blind Week 34- Tapering Arm | 3.0 (3.29) | 0.2 (1.17)
  Double Blind Week 34- Withdrawal Arm: number analyzed (Participants) | 2 | 11
  Double Blind Week 34- Withdrawal Arm | 0.1 (0.33) | 0.1 (1.07)
  Double Blind Week 40- Tapering Arm: number analyzed (Participants) | 11 | 63
  Double Blind Week 40- Tapering Arm | 7.5 (10.27) | 0.1 (1.37)
  Double Blind Week 40- Withdrawal Arm: number analyzed (Participants) | 2 | 11
  Double Blind Week 40- Withdrawal Arm | 8.5 (10.23) | -0.3 (0.62)
  Flare Week 0- Tapering Arm: number analyzed (Participants) | 30 | 0
  Flare Week 0- Tapering Arm | 11.6 (11.17) |
  Flare Week 0- Withdrawal Arm: number analyzed (Participants) | 8 | 0
  Flare Week 0- Withdrawal Arm | 9.9 (8.31) |
  Flare Week 4- Tapering Arm: number analyzed (Participants) | 28 | 0
  Flare Week 4- Tapering Arm | 4.1 (8.73) |
  Flare Week 4- Withdrawal Arm: number analyzed (Participants) | 7 | 0
  Flare Week 4- Withdrawal Arm | 5.2 (9.64) |
  Flare Week 10- Tapering Arm: number analyzed (Participants) | 29 | 0
  Flare Week 10- Tapering Arm | 2.5 (7.53) |
  Flare Week 10- Withdrawal Arm: number analyzed (Participants) | 7 | 0
  Flare Week 10- Withdrawal Arm | 3.5 (2.51) |
  Flare Week 16- Tapering Arm: number analyzed (Participants) | 29 | 0
  Flare Week 16- Tapering Arm | 3.6 (6.63) |
  Flare Week 16- Withdrawal Arm: number analyzed (Participants) | 8 | 0
  Flare Week 16- Withdrawal Arm | 2.7 (4.20) |

13. Secondary Outcome: Number of Participants Maintaining Clinical Remission Defined By DAS28 (ESR) < 2.6, SDAI ≤ 3.3, and CDAI ≤ 2.8 at Each Visit By Treatment Arm
Description: The maintenance of clinical remission after regaining remission during the Open-label rescue period was defined as either Disease Activity Score 28 (DAS28 ESR) < 2.6, Simplified Disease Activity Index (SDAI) score ≤ 3.3, or Clinical Disease Activity Index (CDAI) score ≤ 2.8).
Time Frame: From Week 4 to Week 40 and from Flare Week 0 to Flare Week 16
Population: Double-blind Treated Subject population: participants who received at least 1 dose of study drug during the Double-blind period; last observation carried forward
Measure: Count of Participants; unit: Participants
Groups:
- DAS28 (ESR) < 2.6: Disease Activity Score 28 (DAS28 ESR) < 2.6
- SDAI ≤ 3.3: Simplified Disease Activity Index (SDAI) score ≤ 3.3
- CDAI ≤ 2.8: Clinical Disease Activity Index (CDAI) score ≤ 2.8
Arm/Group | DAS28 (ESR) < 2.6 | SDAI ≤ 3.3 | CDAI ≤ 2.8
Number analyzed (Participants) | 122 | 122 | 122
Participants
  Double Blind Baseline- Tapering Arm: number analyzed (Participants) | 102 | 102 | 102
  Double Blind Baseline- Tapering Arm | 102 | 89 | 85
  Double Blind Baseline- Withdrawal Arm: number analyzed (Participants) | 20 | 20 | 20
  Double Blind Baseline- Withdrawal Arm | 20 | 19 | 19
  Double Blind Week 10- Tapering Arm: number analyzed (Participants) | 100 | 98 | 99
  Double Blind Week 10- Tapering Arm | 85 | 63 | 62
  Double Blind Week 10- Withdrawal Arm: number analyzed (Participants) | 20 | 20 | 20
  Double Blind Week 10- Withdrawal Arm | 18 | 16 | 14
  Double Blind Week 16- Tapering Arm: number analyzed (Participants) | 98 | 98 | 98
  Double Blind Week 16- Tapering Arm | 78 | 64 | 62
  Double Blind Week 16- Withdrawal arm: number analyzed (Participants) | 20 | 20 | 20
  Double Blind Week 16- Withdrawal arm | 15 | 13 | 15
  Double Blind Week 22- Tapering Arm: number analyzed (Participants) | 82 | 82 | 82
  Double Blind Week 22- Tapering Arm | 75 | 59 | 58
  Double Blind Week 22- Withdrawal Arm: number analyzed (Participants) | 15 | 15 | 15
  Double Blind Week 22- Withdrawal Arm | 14 | 13 | 13
  Double Blind Week 28- Tapering Arm: number analyzed (Participants) | 79 | 79 | 79
  Double Blind Week 28- Tapering Arm | 69 | 58 | 57
  Double Blind Week 28- Withdrawal Arm: number analyzed (Participants) | 15 | 15 | 15
  Double Blind Week 28- Withdrawal Arm | 13 | 12 | 13
  Double Blind Week 34- Tapering Arm: number analyzed (Participants) | 75 | 75 | 75
  Double Blind Week 34- Tapering Arm | 70 | 58 | 58
  Double Blind Week 34- Withdrawal Arm: number analyzed (Participants) | 13 | 13 | 13
  Double Blind Week 34- Withdrawal Arm | 13 | 13 | 13
  Double Blind Week 40- Tapering Arm: number analyzed (Participants) | 74 | 74 | 74
  Double Blind Week 40- Tapering Arm | 64 | 57 | 56
  Double Blind Week 40- Withdrawal Arm: number analyzed (Participants) | 13 | 13 | 13
  Double Blind Week 40- Withdrawal Arm | 11 | 12 | 12
  Flare Week 0- Tapering Arm: number analyzed (Participants) | 31 | 31 | 31
  Flare Week 0- Tapering Arm | 4 | 4 | 4
  Flare Week 0- Withdrawal Arm: number analyzed (Participants) | 8 | 8 | 8
  Flare Week 0- Withdrawal Arm | 1 | 0 | 2
  Flare Week 4- Tapering Arm: number analyzed (Participants) | 29 | 28 | 28
  Flare Week 4- Tapering Arm | 14 | 13 | 13
  Flare Week 4- Withdrawal Arm: number analyzed (Participants) | 7 | 7 | 7
  Flare Week 4- Withdrawal Arm | 1 | 2 | 2
  Flare Week 10- Tapering Arm: number analyzed (Participants) | 29 | 29 | 29
  Flare Week 10- Tapering Arm | 17 | 14 | 14
  Flare Week 10- Withdrawal Arm: number analyzed (Participants) | 7 | 7 | 7
  Flare Week 10- Withdrawal Arm | 3 | 2 | 2
  Flare Week 16- Tapering Arm: number analyzed (Participants) | 29 | 29 | 29
  Flare Week 16- Tapering Arm | 13 | 13 | 13
  Flare Week 16- Withdrawal Arm: number analyzed (Participants) | 8 | 8 | 8
  Flare Week 16- Withdrawal Arm | 4 | 4 | 4

14. Secondary Outcome: Mean Change From Double-blind Baseline to Week 40 or Final Visit in Magnetic Resonance Imaging (MRI) Synovitis Score
Description: Synovitis was assessed in three wrist regions (the distal radioulnar joint; the radiocarpal joint; the intercarpal and carpometacarpal joints) and in each Metacarpophalangeal joint (MCP) joint. The first carpometacarpal joint and the first MCP joint are not scored. The scale is 0-3. Score 0 is normal, and 1-3 (mild, moderate, severe) are by thirds of the presumed maximum volume of enhancing tissue in the synovial compartment.
Time Frame: From Week 4 to Week 40 or Final visit
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Flared Participants | Non-Flared Participants
Number analyzed (Participants) | 45 | 76
units on a scale
  Double Blind Week 40- Tapering Arm: number analyzed (Participants) | 6 | 51
  Double Blind Week 40- Tapering Arm | -0.1 (1.20) | 0.1 (1.33)
  Double Blind Week 40- Withdrawal Arm: number analyzed (Participants) | 1 | 10
  Double Blind Week 40- Withdrawal Arm | 0.0 | -0.1 (0.90)
  Flare Week 16- Tapering Arm: number analyzed (Participants) | 25 | 0
  Flare Week 16- Tapering Arm | 0.8 (1.84) |
  Flare Week 16- Withdrawal Arm: number analyzed (Participants) | 7 | 0
  Flare Week 16- Withdrawal Arm | 0.1 (1.81) |

15. Secondary Outcome: Mean Change From Double-blind Baseline to Week 40 or Final Visit in Bone Marrow Edema (BME) Score
Description: Bone edema in each bone was scored separately. The scale is 0-3 based on the proportion of bone with edema, as follows-0: no edema; 1: 1-33% of bone edematous; 2: 34-66% of bone edematous; 3: 67-100%.
Time Frame: From Week 4 to Week 40 or Final visit
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Flared Participants | Non-Flared Participants
Number analyzed (Participants) | 46 | 76
units on a scale
  Double Blind Week 40- Tapering Arm: number analyzed (Participants) | 6 | 52
  Double Blind Week 40- Tapering Arm | -0.5 (0.84) | 0.0 (1.07)
  Double Blind Week 40- Withdrawal Arm: number analyzed (Participants) | 1 | 10
  Double Blind Week 40- Withdrawal Arm | 0.0 | 1.2 (3.52)
  Flare Week 16- Tapering Arm: number analyzed (Participants) | 26 | 0
  Flare Week 16- Tapering Arm | -0.1 (0.47) |
  Flare Week 16- Withdrawal Arm: number analyzed (Participants) | 8 | 0
  Flare Week 16- Withdrawal Arm | 0.3 (0.38) |

16. Secondary Outcome: Mean Change From Double-blind Baseline to Week 40 or Final Visit in Bone Erosions Rheumatoid Arthritis Magnetic Resonance Imaging Scoring System (RAMRIS) Score
Description: Bone erosions in each bone (wrists: carpal bones, distal radius, distal ulna, metacarpal bases; MCP joints: metacarpal heads, phalangeal bases) were scored separately. The scale is 0-10, based on the proportion of eroded bone compared to the ''assessed bone volume'', judged on all available images-0: no erosion; 1: 1-10% of bone eroded; 2; 11-20%, etc.
Time Frame: From Week 4 to Week 40 or Final Visit
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Flared Participants | Non-Flared Participants
Number analyzed (Participants) | 46 | 76
units on a scale
  Double Blind Week 40- Tapering Arm: number analyzed (Participants) | 6 | 52
  Double Blind Week 40- Tapering Arm | -0.5 (1.73) | 0.1 (0.52)
  Double Blind Week 40- Withdrawal Arm: number analyzed (Participants) | 1 | 10
  Double Blind Week 40- Withdrawal Arm | -2.0 | 0.0 (1.08)
  Flare Week 16- Tapering Arm: number analyzed (Participants) | 26 | 0
  Flare Week 16- Tapering Arm | 0.3 (1.02) |
  Flare Week 16- Withdrawal Arm: number analyzed (Participants) | 8 | 0
  Flare Week 16- Withdrawal Arm | 0.1 (0.88) |

17. Secondary Outcome: Mean Change From Double-blind Baseline in Health Assessment Questionnaire- Disability Index (HAQ-DI) Score Over Time
Description: The Health Assessment Questionnaire - Disability Index (HAQ-DI) is a participant-reported questionnaire specific for rheumatoid arthritis. It consists of 20 questions referring to eight domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and daily activities. Participants assessed their ability to do each task over the past week using the following response categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task were summed and averaged to provide an overall score ranging from 0 to 3, where zero represents no disability and three very severe, high-dependency disability. The minimal clinically important difference (MCID) defined for the HAQ-DI is ≥ 0.22.
Time Frame: From Week 4 to Week 40 and from Flare Week 0 to Flare Week 16
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Flared Participants | Non-Flared Participants
Number analyzed (Participants) | 46 | 76
units on a scale
  Double Blind Week 10- Tapering Arm: number analyzed (Participants) | 30 | 62
  Double Blind Week 10- Tapering Arm | 0.1 (0.3) | 0.0 (0.18)
  Double Blind Week 10- Withdrawal Arm: number analyzed (Participants) | 9 | 11
  Double Blind Week 10- Withdrawal Arm | 0.3 (0.61) | 0.0 (0.17)
  Double Blind Week 16- Tapering Arm: number analyzed (Participants) | 19 | 63
  Double Blind Week 16- Tapering Arm | 0.2 (0.40) | -0.0 (0.28)
  Double Blind Week 16- Withdrawal Arm: number analyzed (Participants) | 5 | 11
  Double Blind Week 16- Withdrawal Arm | 0.3 (0.54) | -0.0 (0.12)
  Double Blind Week 22- Tapering Arm: number analyzed (Participants) | 15 | 63
  Double Blind Week 22- Tapering Arm | 0.1 (0.37) | -0.0 (0.26)
  Double Blind Week 22- Withdrawal Arm: number analyzed (Participants) | 4 | 11
  Double Blind Week 22- Withdrawal Arm | 0.4 (0.79) | 0.1 (0.39)
  Double Blind Week 28- Tapering Arm: number analyzed (Participants) | 12 | 63
  Double Blind Week 28- Tapering Arm | 0.2 (0.43) | -0.0 (0.27)
  Double Blind Week 28- Withdrawal Arm: number analyzed (Participants) | 3 | 11
  Double Blind Week 28- Withdrawal Arm | 0.7 (0.69) | -0.1 (0.15)
  Double Blind Week 34- Tapering Arm: number analyzed (Participants) | 11 | 63
  Double Blind Week 34- Tapering Arm | 0.3 (0.49) | -0.0 (0.30)
  Double Blind Week 34- Withdrawal Arm: number analyzed (Participants) | 2 | 11
  Double Blind Week 34- Withdrawal Arm | 0.2 (0.27) | 0.1 (0.17)
  Double Blind Week 40- Tapering Arm: number analyzed (Participants) | 7 | 63
  Double Blind Week 40- Tapering Arm | 0.4 (0.40) | -0.1 (0.33)
  Double Blind Week 40- Withdrawal Arm: number analyzed (Participants) | 1 | 11
  Double Blind Week 40- Withdrawal Arm | 1.9 | 0.0 (0.16)
  Flare Week 0- Tapering Arm: number analyzed (Participants) | 25 | 0
  Flare Week 0- Tapering Arm | 0.4 (0.57) |
  Flare Week 0- Withdrawal Arm: number analyzed (Participants) | 7 | 0
  Flare Week 0- Withdrawal Arm | 0.3 (0.29) |
  Flare Week 4- Tapering Arm: number analyzed (Participants) | 27 | 0
  Flare Week 4- Tapering Arm | 0.2 (0.49) |
  Flare Week 4- Withdrawal Arm: number analyzed (Participants) | 7 | 0
  Flare Week 4- Withdrawal Arm | 0.2 (0.35) |
  Flare Week 10- Tapering Arm: number analyzed (Participants) | 27 | 0
  Flare Week 10- Tapering Arm | 0.1 (0.24) |
  Flare Week 10- Withdrawal Arm: number analyzed (Participants) | 7 | 0
  Flare Week 10- Withdrawal Arm | 0.1 (0.20) |
  Flare Week 16- Tapering Arm: number analyzed (Participants) | 29 | 0
  Flare Week 16- Tapering Arm | 0.2 (0.39) |
  Flare Week 16- Withdrawal Arm: number analyzed (Participants) | 7 | 0
  Flare Week 16- Withdrawal Arm | 0.1 (0.24) |

18. Secondary Outcome: Number of Participants With Health Assessment Questionnaire- Disability Index (HAQ-DI) Score ≤ 0.5 at Double-blind Baseline and at Week 40
Description: The Health Assessment Questionnaire - Disability Index (HAQ-DI) is a participant-reported questionnaire specific for rheumatoid arthritis. It consists of 20 questions referring to eight domains: dressing/grooming, arising, eating, walking, hygiene, reach, grip, and daily activities. Participants assessed their ability to do each task over the past week using the following response categories: without any difficulty (0); with some difficulty (1); with much difficulty (2); and unable to do (3). Scores on each task were summed and averaged to provide an overall score ranging from 0 to 3, where zero represents no disability and three very severe, high-dependency disability. The number of participants with HAQ-DI score ≤ 0.5 (considered to be normal) was recorded.
Time Frame: Week 4 and Week 40
Population: as for outcome 10
Measure: Count of Participants; unit: Participants
Arm/Group | Flared Participants | Non-Flared Participants
Number analyzed (Participants) | 46 | 76
Participants
  Double Blind Week 4- Tapering Arm: number analyzed (Participants) | 37 | 65
  Double Blind Week 4- Tapering Arm | 21 | 50
  Double Blind Week 4- Withdrawal Arm: number analyzed (Participants) | 9 | 11
  Double Blind Week 4- Withdrawal Arm | 7 | 10
  Double Blind Week 40- Tapering Arm: number analyzed (Participants) | 7 | 63
  Double Blind Week 40- Tapering Arm | 2 | 48
  Double Blind Week 40- Withdrawal Arm: number analyzed (Participants) | 1 | 11
  Double Blind Week 40- Withdrawal Arm | 0 | 9

19. Secondary Outcome: Mean Change From Double-blind Baseline in Routine Assessment of Patient Index Data (RAPID3) Questionnaire Scores Assessed During In-office Visits
Description: The RAPID3 is an activity index derived from the Multi-dimensional Health Assessment Questionnaire (MD-HAQ). It includes an assessment of physical function, a pain Visual Analog Scale (VAS), and a participant global assessment of disease activity VAS. The total RAPID3 score ranges from 0 to 30 where higher scores represent severe disease. Negative values indicate improvement from the Double-blind baseline score.
Time Frame: From Week 4 to Week 40 and from Flare Week 0 to Flare Week 16
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Flared Participants | Non-Flared Participants
Number analyzed (Participants) | 46 | 76
units on a scale
  Double Blind Week 10- Tapering Arm: number analyzed (Participants) | 37 | 63
  Double Blind Week 10- Tapering Arm | 1.9 (3.92) | 0.7 (3.20)
  Double Blind Week 10- Withdrawal Arm: number analyzed (Participants) | 9 | 11
  Double Blind Week 10- Withdrawal Arm | 1.4 (3.73) | 1.5 (4.67)
  Double Blind Week 16- Tapering Arm: number analyzed (Participants) | 35 | 63
  Double Blind Week 16- Tapering Arm | 4.7 (5.66) | 0.8 (2.80)
  Double Blind Week 16- Withdrawal Arm: number analyzed (Participants) | 9 | 11
  Double Blind Week 16- Withdrawal Arm | 2.5 (4.59) | 0.1 (1.37)
  Double Blind Week 22- Tapering Arm: number analyzed (Participants) | 19 | 63
  Double Blind Week 22- Tapering Arm | 2.6 (4.83) | 0.3 (2.83)
  Double Blind Week 22- Withdrawal arm: number analyzed (Participants) | 4 | 11
  Double Blind Week 22- Withdrawal arm | 3.6 (4.18) | 0.6 (3.31)
  Double Blind Week 28- Tapering arm: number analyzed (Participants) | 16 | 63
  Double Blind Week 28- Tapering arm | 2.2 (4.20) | 0.6 (2.47)
  Double Blind Week 28- Withdrawal Arm: number analyzed (Participants) | 4 | 11
  Double Blind Week 28- Withdrawal Arm | 3.7 (4.45) | -0.3 (1.61)
  Double Blind Week 34- Tapering Arm: number analyzed (Participants) | 12 | 63
  Double Blind Week 34- Tapering Arm | 2.2 (3.77) | -0.0 (1.93)
  Double Blind Week 34- Withdrawal Arm: number analyzed (Participants) | 2 | 11
  Double Blind Week 34- Withdrawal Arm | 1.9 (2.62) | 1.6 (2.33)
  Double Blind Week 40- Tapering Arm: number analyzed (Participants) | 11 | 63
  Double Blind Week 40- Tapering Arm | 4.7 (6.22) | 0.0 (2.39)
  Double Blind Week 40- Withdrawal Arm: number analyzed (Participants) | 2 | 11
  Double Blind Week 40- Withdrawal Arm | 0.4 (0.92) | 0.8 (1.62)
  Flare Week 0- Tapering Arm: number analyzed (Participants) | 30 | 0
  Flare Week 0- Tapering Arm | 6.1 (6.64) |
  Flare Week 0- Withdrawal Arm: number analyzed (Participants) | 8 | 0
  Flare Week 0- Withdrawal Arm | 3.9 (5.60) |
  Flare Week 4- Tapering Arm: number analyzed (Participants) | 27 | 0
  Flare Week 4- Tapering Arm | 3.1 (5.38) |
  Flare Week 4- Withdrawal Arm: number analyzed (Participants) | 7 | 0
  Flare Week 4- Withdrawal Arm | 3.2 (4.15) |
  Flare Week 10- Tapering Arm: number analyzed (Participants) | 27 | 0
  Flare Week 10- Tapering Arm | 2.8 (3.93) |
  Flare Week 10- Withdrawal Arm: number analyzed (Participants) | 7 | 0
  Flare Week 10- Withdrawal Arm | 2.3 (2.61) |
  Flare Week 16- Tapering Arm: number analyzed (Participants) | 29 | 0
  Flare Week 16- Tapering Arm | 2.9 (4.22) |
  Flare Week 16- Withdrawal Arm: number analyzed (Participants) | 7 | 0
  Flare Week 16- Withdrawal Arm | 2.1 (3.01) |

20. Secondary Outcome: Mean Change From Flare Week 0 in Routine Assessment of Patient Index Data (RAPID3) Questionnaire Scores Assessed at Home
Description: as for outcome 19
Time Frame: Flare Week 0 and Flare Weeks 1, 2, 3, 5, 6, 7, 8, 9, 11, 12, 13, 14, 15
Population: All Open-label rescue treated participants with available data; last observation carried forward
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Flared Participants
Number analyzed (Participants) | 33
units on a scale
  Flare Week 1- Tapering Arm: number analyzed (Participants) | 19
  Flare Week 1- Tapering Arm | -1.6 (4.92)
  Flare Week 1- Withdrawal Arm: number analyzed (Participants) | 3
  Flare Week 1- Withdrawal Arm | 3.7 (7.20)
  Flare Week 2- Tapering Arm: number analyzed (Participants) | 22
  Flare Week 2- Tapering Arm | -3.1 (5.41)
  Flare Week 2- Withdrawal Arm: number analyzed (Participants) | 4
  Flare Week 2- Withdrawal Arm | 0.8 (6.89)
  Flare Week 3- Tapering Arm: number analyzed (Participants) | 25
  Flare Week 3- Tapering Arm | -3.8 (6.78)
  Flare Week 3- Withdrawal Arm: number analyzed (Participants) | 6
  Flare Week 3- Withdrawal Arm | -0.4 (7.94)
  Flare Week 5- Tapering Arm: number analyzed (Participants) | 26
  Flare Week 5- Tapering Arm | -3.8 (6.61)
  Flare Week 5- Withdrawal Arm: number analyzed (Participants) | 6
  Flare Week 5- Withdrawal Arm | -0.8 (6.56)
  Flare Week 6- Tapering Arm: number analyzed (Participants) | 26
  Flare Week 6- Tapering Arm | -4.1 (6.81)
  Flare Week 6- Withdrawal Arm: number analyzed (Participants) | 6
  Flare Week 6- Withdrawal Arm | -0.9 (6.97)
  Flare Week 7- Tapering Arm: number analyzed (Participants) | 26
  Flare Week 7- Tapering Arm | -3.7 (6.86)
  Flare Week 7- Withdrawal Arm: number analyzed (Participants) | 6
  Flare Week 7- Withdrawal Arm | -0.6 (6.26)
  Flare Week 8- Tapering Arm: number analyzed (Participants) | 27
  Flare Week 8- Tapering Arm | -4.4 (7.17)
  Flare Week 8- Withdrawal Arm: number analyzed (Participants) | 6
  Flare Week 8- Withdrawal Arm | -0.6 (5.56)
  Flare Week 9- Tapering Arm: number analyzed (Participants) | 27
  Flare Week 9- Tapering Arm | -3.3 (5.81)
  Flare Week 9- Withdrawal Arm: number analyzed (Participants) | 6
  Flare Week 9- Withdrawal Arm | -1.0 (5.89)
  Flare Week 11- Tapering Arm: number analyzed (Participants) | 27
  Flare Week 11- Tapering Arm | -3.7 (5.69)
  Flare Week 11- Withdrawal Arm: number analyzed (Participants) | 6
  Flare Week 11- Withdrawal Arm | -1.0 (5.85)
  Flare Week 12- Tapering Arm: number analyzed (Participants) | 27
  Flare Week 12- Tapering Arm | -3.4 (5.84)
  Flare Week 12- Withdrawal Arm: number analyzed (Participants) | 6
  Flare Week 12- Withdrawal Arm | -2.3 (4.46)
  Flare Week 13- Tapering Arm: number analyzed (Participants) | 27
  Flare Week 13- Tapering Arm | -3.5 (5.72)
  Flare Week 13- Withdrawal Arm: number analyzed (Participants) | 6
  Flare Week 13- Withdrawal Arm | -2.5 (4.78)
  Flare Week 14- Tapering Arm: number analyzed (Participants) | 27
  Flare Week 14- Tapering Arm | -3.1 (5.54)
  Flare Week 14- Withdrawal Arm: number analyzed (Participants) | 6
  Flare Week 14- Withdrawal Arm | -2.4 (4.79)
  Flare Week 15- Tapering Arm: number analyzed (Participants) | 27
  Flare Week 15- Tapering Arm | -3.5 (6.69)
  Flare Week 15- Withdrawal Arm: number analyzed (Participants) | 6
  Flare Week 15- Withdrawal Arm | -2.2 (4.70)

21. Secondary Outcome: Mean Change From Double-blind Baseline in Swollen Joint Count 28
Description: Twenty-eight joints, excluding hip joints, were assessed for swelling by physical examination. Swelling of each joint was classified as present (1) or absent (0), for a total possible score of 0 (0 joints with swelling) to 28 (worst possible score/28 joints with swelling). Negative values indicate improvement from baseline.
Time Frame: From Week 4 to Week 40 and from Flare Week 0 to Flare Week 16
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: swollen joint counts
Arm/Group | Flared Participants | Non-Flared Participants
Number analyzed (Participants) | 46 | 76
swollen joint counts
  Double Blind Week 10- Tapering Arm: number analyzed (Participants) | 37 | 64
  Double Blind Week 10- Tapering Arm | 0.9 (2.09) | 0.1 (0.58)
  Double Blind Week 10- Withdrawal Arm: number analyzed (Participants) | 9 | 11
  Double Blind Week 10- Withdrawal Arm | 0.1 (0.33) | -0.1 (0.30)
  Double Blind Week 16- Tapering Arm: number analyzed (Participants) | 35 | 63
  Double Blind Week 16- Tapering Arm | 1.2 (2.15) | -0.0 (0.34)
  Double Blind Week 16- Withdrawal Arm: number analyzed (Participants) | 9 | 11
  Double Blind Week 16- Withdrawal Arm | 0.3 (0.50) | 0.0 (0.45)
  Double Blind Week 22- Tapering Arm: number analyzed (Participants) | 19 | 63
  Double Blind Week 22- Tapering Arm | 0.6 (1.64) | 0.1 (0.64)
  Double Blind Week 22- Withdrawal arm: number analyzed (Participants) | 4 | 11
  Double Blind Week 22- Withdrawal arm | 0.5 (0.58) | -0.1 (0.30)
  Double Blind Week 28- Tapering arm: number analyzed (Participants) | 16 | 63
  Double Blind Week 28- Tapering arm | 0.5 (0.89) | 0.0 (0.33)
  Double Blind Week 28- Withdrawal Arm: number analyzed (Participants) | 4 | 11
  Double Blind Week 28- Withdrawal Arm | 2.0 (2.45) | -0.1 (0.30)
  Double Blind Week 34- Tapering Arm: number analyzed (Participants) | 12 | 63
  Double Blind Week 34- Tapering Arm | 0.0 (0.43) | 0.0 (0.46)
  Double Blind Week 34- Withdrawal Arm: number analyzed (Participants) | 2 | 11
  Double Blind Week 34- Withdrawal Arm | 0.0 (0.00) | -0.1 (0.30)
  Double Blind Week 40- Tapering Arm: number analyzed (Participants) | 11 | 63
  Double Blind Week 40- Tapering Arm | 1.5 (3.01) | 0.0 (0.42)
  Double Blind Week 40- Withdrawal Arm: number analyzed (Participants) | 2 | 11
  Double Blind Week 40- Withdrawal Arm | 2.0 (2.83) | -0.1 (0.30)
  Flare Week 0- Tapering Arm: number analyzed (Participants) | 30 | 0
  Flare Week 0- Tapering Arm | 2.3 (2.60) |
  Flare Week 0- Withdrawal Arm: number analyzed (Participants) | 8 | 0
  Flare Week 0- Withdrawal Arm | 1.9 (2.10) |
  Flare Week 4- Tapering Arm: number analyzed (Participants) | 30 | 0
  Flare Week 4- Tapering Arm | 1.2 (1.98) |
  Flare Week 4- Withdrawal Arm: number analyzed (Participants) | 8 | 0
  Flare Week 4- Withdrawal Arm | 0.6 (1.06) |
  Flare Week 10- Tapering Arm: number analyzed (Participants) | 30 | 0
  Flare Week 10- Tapering Arm | 0.4 (0.89) |
  Flare Week 10- Withdrawal Arm: number analyzed (Participants) | 8 | 0
  Flare Week 10- Withdrawal Arm | 0.1 (0.35) |
  Flare Week 16- Tapering Arm: number analyzed (Participants) | 30 | 0
  Flare Week 16- Tapering Arm | 0.9 (1.81) |
  Flare Week 16- Withdrawal Arm: number analyzed (Participants) | 8 | 0
  Flare Week 16- Withdrawal Arm | 0.3 (0.46) |

22. Secondary Outcome: Mean Change From Double-blind Baseline in Swollen Joint Count 66
Description: Sixty-six joints were assessed for swelling by physical examination. Swelling of each joint was classified as present (1) or absent (0), for a total possible score of 0 (0 joints with swelling) to 66 (worst possible score/66 joints with swelling). Negative values indicate improvement from baseline.
Time Frame: From Week 4 to Week 40 and from Flare Week 0 to Flare Week 16
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: swollen joint counts
Arm/Group | Flared Participants | Non-Flared Participants
Number analyzed (Participants) | 46 | 76
swollen joint counts
  Double Blind Week 10- Tapering Arm: number analyzed (Participants) | 37 | 64
  Double Blind Week 10- Tapering Arm | 1.1 (2.36) | 0.1 (0.67)
  Double Blind Week 10- Withdrawal Arm: number analyzed (Participants) | 9 | 11
  Double Blind Week 10- Withdrawal Arm | 0.1 (0.33) | -0.2 (0.40)
  Double Blind Week 16- Tapering Arm: number analyzed (Participants) | 35 | 63
  Double Blind Week 16- Tapering Arm | 1.4 (2.56) | -0.0 (0.34)
  Double Blind Week 16- Withdrawal Arm: number analyzed (Participants) | 9 | 11
  Double Blind Week 16- Withdrawal Arm | 0.4 (0.53) | 0.0 (0.45)
  Double Blind Week 22- Tapering Arm: number analyzed (Participants) | 19 | 63
  Double Blind Week 22- Tapering Arm | 0.6 (1.64) | 0.1 (0.73)
  Double Blind Week 22- Withdrawal arm: number analyzed (Participants) | 4 | 11
  Double Blind Week 22- Withdrawal arm | 1.0 (1.41) | -0.1 (0.30)
  Double Blind Week 28- Tapering arm: number analyzed (Participants) | 16 | 63
  Double Blind Week 28- Tapering arm | 0.5 (0.89) | 0.1 (0.66)
  Double Blind Week 28- Withdrawal Arm: number analyzed (Participants) | 4 | 11
  Double Blind Week 28- Withdrawal Arm | 3.3 (4.72) | -0.2 (0.40)
  Double Blind Week 34- Tapering Arm: number analyzed (Participants) | 12 | 63
  Double Blind Week 34- Tapering Arm | 0.0 (0.43) | 0.0 (0.54)
  Double Blind Week 34- Withdrawal Arm: number analyzed (Participants) | 2 | 11
  Double Blind Week 34- Withdrawal Arm | 0.0 (0.00) | -0.2 (0.40)
  Double Blind Week 40- Tapering Arm: number analyzed (Participants) | 11 | 63
  Double Blind Week 40- Tapering Arm | 1.5 (3.01) | 0.0 (0.46)
  Double Blind Week 40- Withdrawal Arm: number analyzed (Participants) | 2 | 11
  Double Blind Week 40- Withdrawal Arm | 2.0 (2.83) | -0.2 (0.40)
  Flare Week 0- Tapering Arm: number analyzed (Participants) | 30 | 0
  Flare Week 0- Tapering Arm | 2.6 (2.90) |
  Flare Week 0- Withdrawal Arm: number analyzed (Participants) | 8 | 0
  Flare Week 0- Withdrawal Arm | 2.6 (3.38) |
  Flare Week 4- Tapering Arm: number analyzed (Participants) | 30 | 0
  Flare Week 4- Tapering Arm | 1.3 (1.99) |
  Flare Week 4- Withdrawal Arm: number analyzed (Participants) | 8 | 0
  Flare Week 4- Withdrawal Arm | 0.6 (1.06) |
  Flare Week 10- Tapering Arm: number analyzed (Participants) | 30 | 0
  Flare Week 10- Tapering Arm | 0.6 (1.10) |
  Flare Week 10- Withdrawal Arm: number analyzed (Participants) | 8 | 0
  Flare Week 10- Withdrawal Arm | 0.4 (0.52) |
  Flare Week 16- Tapering Arm: number analyzed (Participants) | 30 | 0
  Flare Week 16- Tapering Arm | 1.1 (2.21) |
  Flare Week 16- Withdrawal Arm: number analyzed (Participants) | 8 | 0
  Flare Week 16- Withdrawal Arm | 0.4 (0.74) |

23. Secondary Outcome: Mean Change From Double-blind Baseline in Tender Joint Count 28
Description: Twenty-eight joints were assessed for tenderness by physical examination. Pain or tenderness of each joint was classified as present (1) or absent (0), for a total possible score of 0 (0 joints with tenderness) to 28 (worst possible score/28 joints with tenderness). Negative values indicate improvement from baseline.
Time Frame: From Week 4 to Week 40 and from Flare Week 0 to Flare Week 16
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: tender joint counts
Arm/Group | Flared Participants | Non-Flared Participants
Number analyzed (Participants) | 46 | 76
tender joint counts
  Double Blind Week 10- Tapering Arm: number analyzed (Participants) | 37 | 64
  Double Blind Week 10- Tapering Arm | 1.3 (2.74) | 0.1 (0.54)
  Double Blind Week 10- Withdrawal Arm: number analyzed (Participants) | 9 | 11
  Double Blind Week 10- Withdrawal Arm | -0.1 (0.60) | 0.5 (1.21)
  Double Blind Week 16- Tapering Arm: number analyzed (Participants) | 35 | 63
  Double Blind Week 16- Tapering Arm | 2.5 (4.49) | 0.1 (0.41)
  Double Blind Week 16- Withdrawal Arm: number analyzed (Participants) | 9 | 11
  Double Blind Week 16- Withdrawal Arm | 1.0 (0.87) | 0.0 (0.00)
  Double Blind Week 22- Tapering Arm: number analyzed (Participants) | 19 | 63
  Double Blind Week 22- Tapering Arm | 0.9 (1.66) | -0.0 (0.42)
  Double Blind Week 22- Withdrawal arm: number analyzed (Participants) | 4 | 11
  Double Blind Week 22- Withdrawal arm | 0.8 (1.50) | 0.1 (0.30)
  Double Blind Week 28- Tapering arm: number analyzed (Participants) | 16 | 63
  Double Blind Week 28- Tapering arm | 1.6 (3.39) | 0.0 (0.51)
  Double Blind Week 28- Withdrawal Arm: number analyzed (Participants) | 4 | 11
  Double Blind Week 28- Withdrawal Arm | 1.8 (2.36) | 0.2 (0.40)
  Double Blind Week 34- Tapering Arm: number analyzed (Participants) | 12 | 63
  Double Blind Week 34- Tapering Arm | 1.0 (1.65) | -0.0 (0.42)
  Double Blind Week 34- Withdrawal Arm: number analyzed (Participants) | 2 | 11
  Double Blind Week 34- Withdrawal Arm | 0.0 (0.00) | 0.0 (0.00)
  Double Blind Week 40- Tapering Arm: number analyzed (Participants) | 11 | 63
  Double Blind Week 40- Tapering Arm | 2.0 (2.65) | 0.0 (0.51)
  Double Blind Week 40- Withdrawal Arm: number analyzed (Participants) | 2 | 11
  Double Blind Week 40- Withdrawal Arm | 3.5 (4.95) | 0.0 (0.00)
  Flare Week 0- Tapering Arm: number analyzed (Participants) | 30 | 0
  Flare Week 0- Tapering Arm | 4.4 (4.63) |
  Flare Week 0- Withdrawal Arm: number analyzed (Participants) | 8 | 0
  Flare Week 0- Withdrawal Arm | 3.6 (3.81) |
  Flare Week 4- Tapering Arm: number analyzed (Participants) | 30 | 0
  Flare Week 4- Tapering Arm | 1.5 (2.27) |
  Flare Week 4- Withdrawal Arm: number analyzed (Participants) | 8 | 0
  Flare Week 4- Withdrawal Arm | 2.5 (5.13) |
  Flare Week 10- Tapering Arm: number analyzed (Participants) | 30 | 0
  Flare Week 10- Tapering Arm | 0.9 (1.84) |
  Flare Week 10- Withdrawal Arm: number analyzed (Participants) | 8 | 0
  Flare Week 10- Withdrawal Arm | 1.1 (1.46) |
  Flare Week 16- Tapering Arm: number analyzed (Participants) | 30 | 0
  Flare Week 16- Tapering Arm | 1.8 (2.64) |
  Flare Week 16- Withdrawal Arm: number analyzed (Participants) | 8 | 0
  Flare Week 16- Withdrawal Arm | 1.1 (1.89) |

24. Secondary Outcome: Mean Change From Double-blind Baseline in Tender Joint Count 68
Description: Sixty-eight joints were assessed for tenderness by physical examination. Pain or tenderness of each joint was classified as present (1) or absent (0), for a total possible score of 0 (0 joints with tenderness) to 68 (worst possible score/68 joints with tenderness). Negative values indicate improvement from baseline.
Time Frame: From Week 4 to Week 40 and from Flare Week 0 to Flare Week 16
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: tender joint counts
Arm/Group | Flared Participants | Non-Flared Participants
Number analyzed (Participants) | 46 | 76
tender joint counts
  Double Blind Week 10- Tapering Arm: number analyzed (Participants) | 37 | 64
  Double Blind Week 10- Tapering Arm | 1.9 (3.45) | 0.3 (1.47)
  Double Blind Week 10- Withdrawal Arm: number analyzed (Participants) | 9 | 11
  Double Blind Week 10- Withdrawal Arm | 0.1 (0.60) | 0.9 (1.64)
  Double Blind Week 16- Tapering Arm: number analyzed (Participants) | 35 | 63
  Double Blind Week 16- Tapering Arm | 3.5 (6.33) | 0.2 (1.36)
  Double Blind Week 16- Withdrawal Arm: number analyzed (Participants) | 9 | 11
  Double Blind Week 16- Withdrawal Arm | 1.4 (1.13) | 0.2 (0.60)
  Double Blind Week 22- Tapering Arm: number analyzed (Participants) | 19 | 63
  Double Blind Week 22- Tapering Arm | 1.2 (2.27) | 0.2 (1.35)
  Double Blind Week 22- Withdrawal arm: number analyzed (Participants) | 4 | 11
  Double Blind Week 22- Withdrawal arm | 2.0 (2.83) | 0.4 (1.03)
  Double Blind Week 28- Tapering arm: number analyzed (Participants) | 16 | 63
  Double Blind Week 28- Tapering arm | 2.5 (5.34) | 0.1 (0.96)
  Double Blind Week 28- Withdrawal Arm: number analyzed (Participants) | 4 | 11
  Double Blind Week 28- Withdrawal Arm | 3.8 (4.50) | 0.3 (0.47)
  Double Blind Week 34- Tapering Arm: number analyzed (Participants) | 12 | 63
  Double Blind Week 34- Tapering Arm | 1.9 (2.87) | 0.0 (0.73)
  Double Blind Week 34- Withdrawal Arm: number analyzed (Participants) | 2 | 11
  Double Blind Week 34- Withdrawal Arm | 0.0 (0.00) | 0.1 (0.30)
  Double Blind Week 40- Tapering Arm: number analyzed (Participants) | 11 | 63
  Double Blind Week 40- Tapering Arm | 3.0 (4.24) | 0.0 (0.68)
  Double Blind Week 40- Withdrawal Arm: number analyzed (Participants) | 2 | 11
  Double Blind Week 40- Withdrawal Arm | 9.0 (12.73) | -0.1 (0.30)
  Flare Week 0- Tapering Arm: number analyzed (Participants) | 30 | 0
  Flare Week 0- Tapering Arm | 6.2 (6.93) |
  Flare Week 0- Withdrawal Arm: number analyzed (Participants) | 8 | 0
  Flare Week 0- Withdrawal Arm | 6.1 (6.27) |
  Flare Week 4- Tapering Arm: number analyzed (Participants) | 30 | 0
  Flare Week 4- Tapering Arm | 1.9 (2.50) |
  Flare Week 4- Withdrawal Arm: number analyzed (Participants) | 8 | 0
  Flare Week 4- Withdrawal Arm | 4.1 (8.48) |
  Flare Week 10- Tapering Arm: number analyzed (Participants) | 30 | 0
  Flare Week 10- Tapering Arm | 1.5 (2.69) |
  Flare Week 10- Withdrawal Arm: number analyzed (Participants) | 8 | 0
  Flare Week 10- Withdrawal Arm | 2.3 (2.31) |
  Flare Week 16- Tapering Arm: number analyzed (Participants) | 30 | 0
  Flare Week 16- Tapering Arm | 2.1 (3.37) |
  Flare Week 16- Withdrawal Arm: number analyzed (Participants) | 8 | 0
  Flare Week 16- Withdrawal Arm | 1.6 (1.85) |

25. Secondary Outcome: Mean Change From Double-blind Baseline in Participant's Global Assessment of Disease Activity
Description: Participants rated the severity of their rheumatoid arthritis symptoms and how well they were doing during the last 24 hours by placing a vertical mark on a line with a range of 0 (very well) to 100 mm (very poorly). Negative values indicate improvement from baseline.
Time Frame: From Week 4 to Week 40 and from Flare Week 0 to Flare Week 16
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Flared Participants | Non-Flared Participants
Number analyzed (Participants) | 46 | 76
units on a scale
  Double Blind Week 10- Tapering Arm: number analyzed (Participants) | 37 | 63
  Double Blind Week 10- Tapering Arm | 11.6 (19.00) | 2.6 (8.49)
  Double Blind Week 10- Withdrawal Arm: number analyzed (Participants) | 9 | 11
  Double Blind Week 10- Withdrawal Arm | 8.0 (21.66) | 9.6 (20.27)
  Double Blind Week 16- Tapering Arm: number analyzed (Participants) | 35 | 63
  Double Blind Week 16- Tapering Arm | 20.5 (26.97) | 2.4 (9.27)
  Double Blind Week 16- Withdrawal Arm: number analyzed (Participants) | 9 | 11
  Double Blind Week 16- Withdrawal Arm | 10.7 (19.97) | -0.3 (5.76)
  Double Blind Week 22- Tapering Arm: number analyzed (Participants) | 19 | 63
  Double Blind Week 22- Tapering Arm | 10.7 (17.74) | 1.7 (9.14)
  Double Blind Week 22- Withdrawal arm: number analyzed (Participants) | 4 | 11
  Double Blind Week 22- Withdrawal arm | 5.8 (8.73) | 0.2 (8.87)
  Double Blind Week 28- Tapering arm: number analyzed (Participants) | 16 | 63
  Double Blind Week 28- Tapering arm | 9.4 (21.03) | 2.7 (10.03)
  Double Blind Week 28- Withdrawal Arm: number analyzed (Participants) | 4 | 11
  Double Blind Week 28- Withdrawal Arm | 15.0 (25.76) | -1.0 (7.82)
  Double Blind Week 34- Tapering Arm: number analyzed (Participants) | 12 | 63
  Double Blind Week 34- Tapering Arm | 11.5 (13.70) | 1.2 (7.23)
  Double Blind Week 34- Withdrawal Arm: number analyzed (Participants) | 2 | 11
  Double Blind Week 34- Withdrawal Arm | -1.0 (1.41) | 0.7 (7.25)
  Double Blind Week 40- Tapering Arm: number analyzed (Participants) | 11 | 63
  Double Blind Week 40- Tapering Arm | 22.9 (35.32) | 0.0 (7.60)
  Double Blind Week 40- Withdrawal Arm: number analyzed (Participants) | 2 | 11
  Double Blind Week 40- Withdrawal Arm | 2.0 (9.90) | -1.7 (4.45)
  Flare Week 0- Tapering Arm: number analyzed (Participants) | 30 | 0
  Flare Week 0- Tapering Arm | 29.5 (29.43) |
  Flare Week 0- Withdrawal Arm: number analyzed (Participants) | 8 | 0
  Flare Week 0- Withdrawal Arm | 21.6 (27.07) |
  Flare Week 4- Tapering Arm: number analyzed (Participants) | 29 | 0
  Flare Week 4- Tapering Arm | 13.7 (22.93) |
  Flare Week 4- Withdrawal Arm: number analyzed (Participants) | 7 | 0
  Flare Week 4- Withdrawal Arm | 11.7 (21.96) |
  Flare Week 10- Tapering Arm: number analyzed (Participants) | 29 | 0
  Flare Week 10- Tapering Arm | 11.7 (16.89) |
  Flare Week 10- Withdrawal Arm: number analyzed (Participants) | 7 | 0
  Flare Week 10- Withdrawal Arm | 14.1 (10.35) |
  Flare Week 16- Tapering Arm: number analyzed (Participants) | 29 | 0
  Flare Week 16- Tapering Arm | 9.4 (13.47) |
  Flare Week 16- Withdrawal Arm: number analyzed (Participants) | 8 | 0
  Flare Week 16- Withdrawal Arm | 6.9 (9.31) |

26. Secondary Outcome: Mean Change From Double-blind Baseline in Participant's Global Assessment of Rheumatoid Arthritis Pain
Description: Participants rated the severity of their rheumatoid arthritis pain in the past week by placing a vertical mark on a line with a range of 0 (no pain) to 100 mm (severe pain). Negative values indicate improvement from baseline.
Time Frame: From Week 4 to Week 40 and from Flare Week 0 to Flare Week 16
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Flared Participants | Non-Flared Participants
Number analyzed (Participants) | 46 | 76
units on a scale
  Double Blind Week 10- Tapering Arm: number analyzed (Participants) | 37 | 63
  Double Blind Week 10- Tapering Arm | 8.0 (17.96) | 3.5 (14.33)
  Double Blind Week 10- Withdrawal Arm: number analyzed (Participants) | 9 | 11
  Double Blind Week 10- Withdrawal Arm | 6.4 (19.05) | 9.3 (21.04)
  Double Blind Week 16- Tapering Arm: number analyzed (Participants) | 35 | 63
  Double Blind Week 16- Tapering Arm | 17.8 (27.16) | 3.0 (12.48)
  Double Blind Week 16- Withdrawal Arm: number analyzed (Participants) | 9 | 11
  Double Blind Week 16- Withdrawal Arm | 10.7 (18.93) | -0.6 (9.65)
  Double Blind Week 22- Tapering Arm: number analyzed (Participants) | 19 | 63
  Double Blind Week 22- Tapering Arm | 10.4 (19.55) | 0.3 (7.82)
  Double Blind Week 22- Withdrawal arm: number analyzed (Participants) | 4 | 11
  Double Blind Week 22- Withdrawal arm | 4.0 (4.90) | -1.1 (11.20)
  Double Blind Week 28- Tapering arm: number analyzed (Participants) | 16 | 63
  Double Blind Week 28- Tapering arm | 8.3 (17.57) | 1.6 (9.83)
  Double Blind Week 28- Withdrawal Arm: number analyzed (Participants) | 4 | 11
  Double Blind Week 28- Withdrawal Arm | 14.0 (24.59) | -1.4 (10.93)
  Double Blind Week 34- Tapering Arm: number analyzed (Participants) | 12 | 63
  Double Blind Week 34- Tapering Arm | 11.6 (14.61) | -0.3 (7.61)
  Double Blind Week 34- Withdrawal Arm: number analyzed (Participants) | 2 | 11
  Double Blind Week 34- Withdrawal Arm | -3.5 (2.12) | 2.1 (8.40)
  Double Blind Week 40- Tapering Arm: number analyzed (Participants) | 11 | 63
  Double Blind Week 40- Tapering Arm | 24.0 (32.67) | -0.5 (10.00)
  Double Blind Week 40- Withdrawal Arm: number analyzed (Participants) | 2 | 11
  Double Blind Week 40- Withdrawal Arm | -0.5 (20.51) | -0.9 (5.07)
  Flare Week 0- Tapering Arm: number analyzed (Participants) | 30 | 0
  Flare Week 0- Tapering Arm | 24.4 (31.66) |
  Flare Week 0- Withdrawal Arm: number analyzed (Participants) | 8 | 0
  Flare Week 0- Withdrawal Arm | 17.0 (19.38) |
  Flare Week 4- Tapering Arm: number analyzed (Participants) | 29 | 0
  Flare Week 4- Tapering Arm | 9.0 (21.68) |
  Flare Week 4- Withdrawal Arm: number analyzed (Participants) | 7 | 0
  Flare Week 4- Withdrawal Arm | 11.1 (17.46) |
  Flare Week 10- Tapering Arm: number analyzed (Participants) | 29 | 0
  Flare Week 10- Tapering Arm | 7.5 (14.93) |
  Flare Week 10- Withdrawal Arm: number analyzed (Participants) | 7 | 0
  Flare Week 10- Withdrawal Arm | 8.3 (9.60) |
  Flare Week 16- Tapering Arm: number analyzed (Participants) | 29 | 0
  Flare Week 16- Tapering Arm | 8.0 (14.41) |
  Flare Week 16- Withdrawal Arm: number analyzed (Participants) | 8 | 0
  Flare Week 16- Withdrawal Arm | 4.3 (6.32) |

27. Secondary Outcome: Mean Change From Double-blind Baseline in Physician's Global Assessment of Disease Activity
Description: Physicians assessed participants' current rheumatoid arthritis disease activity at the time of the visit (independent of the participant's self-assessment) by placing a vertical mark on a line with a range of 0 (very low) to 100 mm (very high). Negative values indicate improvement from baseline.
Time Frame: From Week 4 to Week 40 and from Flare Week 0 to Flare Week 16
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Flared Participants | Non-Flared Participants
Number analyzed (Participants) | 46 | 76
units on a scale
  Double Blind Week 10- Tapering Arm: number analyzed (Participants) | 37 | 62
  Double Blind Week 10- Tapering Arm | 10.2 (19.54) | 1.3 (4.27)
  Double Blind Week 10- Withdrawal Arm: number analyzed (Participants) | 9 | 11
  Double Blind Week 10- Withdrawal Arm | 1.6 (4.67) | 0.5 (4.74)
  Double Blind Week 16- Tapering Arm: number analyzed (Participants) | 35 | 63
  Double Blind Week 16- Tapering Arm | 13.2 (21.48) | 0.9 (5.07)
  Double Blind Week 16- Withdrawal Arm: number analyzed (Participants) | 9 | 11
  Double Blind Week 16- Withdrawal Arm | 5.0 (3.35) | -0.5 (2.98)
  Double Blind Week 22- Tapering Arm: number analyzed (Participants) | 19 | 63
  Double Blind Week 22- Tapering Arm | 6.9 (14.83) | 0.9 (5.05)
  Double Blind Week 22- Withdrawal arm: number analyzed (Participants) | 4 | 11
  Double Blind Week 22- Withdrawal arm | 3.8 (2.87) | 0.4 (3.26)
  Double Blind Week 28- Tapering arm: number analyzed (Participants) | 16 | 63
  Double Blind Week 28- Tapering arm | 7.3 (16.51) | 1.7 (5.51)
  Double Blind Week 28- Withdrawal Arm: number analyzed (Participants) | 4 | 11
  Double Blind Week 28- Withdrawal Arm | 10.0 (10.89) | -0.9 (2.74)
  Double Blind Week 34- Tapering Arm: number analyzed (Participants) | 12 | 63
  Double Blind Week 34- Tapering Arm | 5.5 (12.27) | 0.8 (3.60)
  Double Blind Week 34- Withdrawal Arm: number analyzed (Participants) | 2 | 11
  Double Blind Week 34- Withdrawal Arm | 0.0 (0.00) | 0.6 (4.13)
  Double Blind Week 40- Tapering Arm: number analyzed (Participants) | 11 | 63
  Double Blind Week 40- Tapering Arm | 16.2 (26.91) | 1.0 (5.32)
  Double Blind Week 40- Withdrawal Arm: number analyzed (Participants) | 2 | 11
  Double Blind Week 40- Withdrawal Arm | 19.5 (26.16) | -0.6 (2.42)
  Flare Week 0- Tapering Arm: number analyzed (Participants) | 30 | 0
  Flare Week 0- Tapering Arm | 26.5 (23.28) |
  Flare Week 0- Withdrawal Arm: number analyzed (Participants) | 8 | 0
  Flare Week 0- Withdrawal Arm | 17.4 (15.37) |
  Flare Week 4- Tapering Arm: number analyzed (Participants) | 29 | 0
  Flare Week 4- Tapering Arm | 12.2 (17.06) |
  Flare Week 4- Withdrawal Arm: number analyzed (Participants) | 7 | 0
  Flare Week 4- Withdrawal Arm | 9.3 (20.27) |
  Flare Week 10- Tapering Arm: number analyzed (Participants) | 30 | 0
  Flare Week 10- Tapering Arm | 10.2 (13.82) |
  Flare Week 10- Withdrawal Arm: number analyzed (Participants) | 7 | 0
  Flare Week 10- Withdrawal Arm | 12.9 (11.51) |
  Flare Week 16- Tapering Arm: number analyzed (Participants) | 30 | 0
  Flare Week 16- Tapering Arm | 8.6 (12.48) |
  Flare Week 16- Withdrawal Arm: number analyzed (Participants) | 8 | 0
  Flare Week 16- Withdrawal Arm | 7.6 (20.00) |

28. Secondary Outcome: Mean Change From Double-blind Baseline in Morning Stiffness Duration
Description: The duration of morning stiffness was reported by participants as the average daily length during the past week in minutes (from time of awaking to time of maximal improvement). Negative values indicate improvement from baseline.
Time Frame: From Week 4 to Week 40 and from Flare Week 0 to Flare Week 16
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Flared Participants | Non-Flared Participants
Number analyzed (Participants) | 45 | 74
minutes
  Double Blind Week 10- Tapering Arm: number analyzed (Participants) | 36 | 62
  Double Blind Week 10- Tapering Arm | 3.5 (17.33) | 1.8 (7.19)
  Double Blind Week 10- Withdrawal Arm: number analyzed (Participants) | 8 | 10
  Double Blind Week 10- Withdrawal Arm | 1.1 (3.60) | 1.5 (5.97)
  Double Blind Week 16- Tapering Arm: number analyzed (Participants) | 34 | 61
  Double Blind Week 16- Tapering Arm | 6.6 (24.41) | 2.3 (12.54)
  Double Blind Week 16- Withdrawal Arm: number analyzed (Participants) | 9 | 11
  Double Blind Week 16- Withdrawal Arm | 9.2 (19.78) | -0.6 (5.05)
  Double Blind Week 22- Tapering Arm: number analyzed (Participants) | 18 | 61
  Double Blind Week 22- Tapering Arm | -1.6 (8.07) | 1.5 (9.67)
  Double Blind Week 22- Withdrawal arm: number analyzed (Participants) | 4 | 11
  Double Blind Week 22- Withdrawal arm | 1.0 (2.00) | 0.5 (3.70)
  Double Blind Week 28- Tapering arm: number analyzed (Participants) | 15 | 61
  Double Blind Week 28- Tapering arm | 2.6 (13.09) | 2.4 (10.53)
  Double Blind Week 28- Withdrawal Arm: number analyzed (Participants) | 4 | 11
  Double Blind Week 28- Withdrawal Arm | 17.3 (28.81) | 0.0 (3.71)
  Double Blind Week 34- Tapering Arm: number analyzed (Participants) | 12 | 61
  Double Blind Week 34- Tapering Arm | 0.6 (10.97) | 1.4 (8.86)
  Double Blind Week 34- Withdrawal Arm: number analyzed (Participants) | 2 | 11
  Double Blind Week 34- Withdrawal Arm | 0.0 (0.00) | -1.1 (6.64)
  Double Blind Week 40- Tapering Arm: number analyzed (Participants) | 11 | 61
  Double Blind Week 40- Tapering Arm | 2.0 (12.49) | 0.4 (9.33)
  Double Blind Week 40- Withdrawal Arm: number analyzed (Participants) | 2 | 11
  Double Blind Week 40- Withdrawal Arm | 0.0 (0.00) | -0.2 (5.78)
  Flare Week 0- Tapering Arm: number analyzed (Participants) | 29 | 0
  Flare Week 0- Tapering Arm | 13.5 (25.21) |
  Flare Week 0- Withdrawal Arm: number analyzed (Participants) | 8 | 0
  Flare Week 0- Withdrawal Arm | 18.5 (26.25) |
  Flare Week 4- Tapering Arm: number analyzed (Participants) | 29 | 0
  Flare Week 4- Tapering Arm | 25.0 (110.77) |
  Flare Week 4- Withdrawal Arm: number analyzed (Participants) | 8 | 0
  Flare Week 4- Withdrawal Arm | 19.9 (26.51) |
  Flare Week 10- Tapering Arm: number analyzed (Participants) | 29 | 0
  Flare Week 10- Tapering Arm | 8.1 (30.20) |
  Flare Week 10- Withdrawal Arm: number analyzed (Participants) | 8 | 0
  Flare Week 10- Withdrawal Arm | 7.9 (9.72) |
  Flare Week 16- Tapering Arm: number analyzed (Participants) | 29 | 0
  Flare Week 16- Tapering Arm | 17.3 (36.46) |
  Flare Week 16- Withdrawal Arm: number analyzed (Participants) | 8 | 0
  Flare Week 16- Withdrawal Arm | 9.6 (20.65) |

29. Secondary Outcome: Mean Change From Double-blind Baseline in Morning Stiffness Severity
Description: Morning stiffness severity was assessed by a numeric rating-scale (NRS). Participants rated the severity of morning stiffness during the past week from 0 to 10 with 0 representing "not severe" and 10 "very severe". Negative values indicate improvement from baseline.
Time Frame: From Week 4 to Week 40 and from Flare Week 0 to Flare Week 16
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Flared Participants | Non-Flared Participants
Number analyzed (Participants) | 46 | 76
units on a scale
  Double Blind Week 10- Tapering Arm: number analyzed (Participants) | 37 | 63
  Double Blind Week 10- Tapering Arm | 0.6 (1.51) | 0.4 (1.01)
  Double Blind Week 10- Withdrawal Arm: number analyzed (Participants) | 9 | 11
  Double Blind Week 10- Withdrawal Arm | 0.4 (1.81) | 0.6 (1.29)
  Double Blind Week 16- Tapering Arm: number analyzed (Participants) | 35 | 63
  Double Blind Week 16- Tapering Arm | 0.8 (1.73) | 0.3 (1.11)
  Double Blind Week 16- Withdrawal Arm: number analyzed (Participants) | 9 | 11
  Double Blind Week 16- Withdrawal Arm | 0.7 (2.24) | -0.1 (1.04)
  Double Blind Week 22- Tapering Arm: number analyzed (Participants) | 19 | 63
  Double Blind Week 22- Tapering Arm | 0.9 (1.27) | 0.2 (0.85)
  Double Blind Week 22- Withdrawal arm: number analyzed (Participants) | 4 | 11
  Double Blind Week 22- Withdrawal arm | 0.8 (0.96) | 0.4 (1.75)
  Double Blind Week 28- Tapering arm: number analyzed (Participants) | 16 | 63
  Double Blind Week 28- Tapering arm | 0.9 (1.69) | 0.2 (1.10)
  Double Blind Week 28- Withdrawal Arm: number analyzed (Participants) | 4 | 11
  Double Blind Week 28- Withdrawal Arm | 1.3 (2.75) | -0.2 (0.87)
  Double Blind Week 34- Tapering Arm: number analyzed (Participants) | 12 | 63
  Double Blind Week 34- Tapering Arm | 1.3 (1.71) | 0.1 (0.85)
  Double Blind Week 34- Withdrawal Arm: number analyzed (Participants) | 2 | 11
  Double Blind Week 34- Withdrawal Arm | 0.0 (1.41) | -0.2 (1.08)
  Double Blind Week 40- Tapering Arm: number analyzed (Participants) | 11 | 63
  Double Blind Week 40- Tapering Arm | 1.8 (2.52) | 0.1 (0.94)
  Double Blind Week 40- Withdrawal Arm: number analyzed (Participants) | 2 | 11
  Double Blind Week 40- Withdrawal Arm | -1.0 (1.41) | -0.4 (1.03)
  Flare Week 0- Tapering Arm: number analyzed (Participants) | 30 | 0
  Flare Week 0- Tapering Arm | 1.6 (2.11) |
  Flare Week 0- Withdrawal Arm: number analyzed (Participants) | 8 | 0
  Flare Week 0- Withdrawal Arm | 0.9 (1.96) |
  Flare Week 4- Tapering Arm: number analyzed (Participants) | 29 | 0
  Flare Week 4- Tapering Arm | 0.8 (2.21) |
  Flare Week 4- Withdrawal Arm: number analyzed (Participants) | 7 | 0
  Flare Week 4- Withdrawal Arm | 0.6 (1.72) |
  Flare Week 10- Tapering Arm: number analyzed (Participants) | 29 | 0
  Flare Week 10- Tapering Arm | 0.6 (1.40) |
  Flare Week 10- Withdrawal Arm: number analyzed (Participants) | 7 | 0
  Flare Week 10- Withdrawal Arm | 0.6 (1.27) |
  Flare Week 16- Tapering Arm: number analyzed (Participants) | 29 | 0
  Flare Week 16- Tapering Arm | 0.6 (1.45) |
  Flare Week 16- Withdrawal Arm: number analyzed (Participants) | 8 | 0
  Flare Week 16- Withdrawal Arm | -0.1 (1.13) |

30. Secondary Outcome: Mean Change From Double-blind Baseline in Participant's Assessment of Sleep Disturbance
Description: Participants rated the severity of their sleep disturbance in the past week by placing a vertical mark on a line with a range of 0 (sleep is no problem) to 100 mm (sleep is a major problem). Negative values indicate improvement from baseline.
Time Frame: From Week 4 to Week 40 and from Flare Week 0 to Flare Week 16
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Flared Participants | Non-Flared Participants
Number analyzed (Participants) | 46 | 76
units on a scale
  Double Blind Week 10- Tapering Arm: number analyzed (Participants) | 37 | 63
  Double Blind Week 10- Tapering Arm | 2.1 (15.37) | 0.0 (8.99)
  Double Blind Week 10- Withdrawal Arm: number analyzed (Participants) | 9 | 11
  Double Blind Week 10- Withdrawal Arm | -3.2 (29.39) | 0.8 (1.54)
  Double Blind Week 16- Tapering Arm: number analyzed (Participants) | 35 | 63
  Double Blind Week 16- Tapering Arm | 10.2 (19.12) | 1.7 (15.96)
  Double Blind Week 16- Withdrawal Arm: number analyzed (Participants) | 9 | 11
  Double Blind Week 16- Withdrawal Arm | 7.1 (22.42) | 1.1 (3.02)
  Double Blind Week 22- Tapering Arm: number analyzed (Participants) | 19 | 63
  Double Blind Week 22- Tapering Arm | 8.2 (19.59) | -0.3 (10.91)
  Double Blind Week 22- Withdrawal arm: number analyzed (Participants) | 4 | 11
  Double Blind Week 22- Withdrawal arm | 8.3 (31.35) | 3.5 (8.70)
  Double Blind Week 28- Tapering arm: number analyzed (Participants) | 16 | 63
  Double Blind Week 28- Tapering arm | 1.8 (27.81) | 2.1 (12.67)
  Double Blind Week 28- Withdrawal Arm: number analyzed (Participants) | 4 | 11
  Double Blind Week 28- Withdrawal Arm | 4.5 (19.82) | -1.0 (7.63)
  Double Blind Week 34- Tapering Arm: number analyzed (Participants) | 12 | 63
  Double Blind Week 34- Tapering Arm | 5.6 (22.99) | -0.4 (11.48)
  Double Blind Week 34- Withdrawal Arm: number analyzed (Participants) | 2 | 11
  Double Blind Week 34- Withdrawal Arm | -0.5 (30.41) | -0.4 (2.77)
  Double Blind Week 40- Tapering Arm: number analyzed (Participants) | 11 | 63
  Double Blind Week 40- Tapering Arm | 17.7 (34.04) | -0.2 (12.40)
  Double Blind Week 40- Withdrawal Arm: number analyzed (Participants) | 2 | 11
  Double Blind Week 40- Withdrawal Arm | -8.0 (15.56) | -1.0 (4.43)
  Flare Week 0- Tapering Arm: number analyzed (Participants) | 30 | 0
  Flare Week 0- Tapering Arm | 18.9 (26.53) |
  Flare Week 0- Withdrawal Arm: number analyzed (Participants) | 8 | 0
  Flare Week 0- Withdrawal Arm | 4.0 (14.61) |
  Flare Week 4- Tapering Arm: number analyzed (Participants) | 29 | 0
  Flare Week 4- Tapering Arm | 4.9 (24.33) |
  Flare Week 4- Withdrawal Arm: number analyzed (Participants) | 7 | 0
  Flare Week 4- Withdrawal Arm | 1.6 (10.05) |
  Flare Week 10- Tapering Arm: number analyzed (Participants) | 29 | 0
  Flare Week 10- Tapering Arm | 0.2 (21.26) |
  Flare Week 10- Withdrawal Arm: number analyzed (Participants) | 7 | 0
  Flare Week 10- Withdrawal Arm | 3.9 (12.98) |
  Flare Week 16- Tapering Arm: number analyzed (Participants) | 29 | 0
  Flare Week 16- Tapering Arm | 2.3 (20.17) |
  Flare Week 16- Withdrawal Arm: number analyzed (Participants) | 8 | 0
  Flare Week 16- Withdrawal Arm | -7.3 (14.14) |

31. Secondary Outcome: Mean Change From Double-blind Baseline in Treatment Satisfaction Questionnaire for Medication (TSQM) Effectiveness Score
Description: Participants completed the 14-item Treatment Satisfaction Questionnaire for Medication (TSQM; Version 1.4) to assess satisfaction with their current rheumatoid arthritis treatment over the previous 2-3 weeks or since the last time that they took the medication. The TSQM consists of fourteen items over four domains (effectiveness, side effects, convenience, and global satisfaction). The 14 questions are answered either with yes/no or by means of a five or seven stage scale (ranging from very unsatisfied to satisfied). TSQM Scale scores for each domain range from 0 to 100 and higher scores represent higher satisfaction. Negative values indicate worsening from baseline.
Time Frame: At Weeks 4, 16, 28, and 40 and from Flare Week 0 to Flare Week 16
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Flared Participants | Non-Flared Participants
Number analyzed (Participants) | 46 | 74
units on a scale
  Double Blind Week 16- Tapering Arm: number analyzed (Participants) | 35 | 61
  Double Blind Week 16- Tapering Arm | -8.3 (35.30) | 0.2 (23.74)
  Double Blind Week 16- Withdrawal Arm: number analyzed (Participants) | 8 | 11
  Double Blind Week 16- Withdrawal Arm | 2.8 (39.51) | -13.6 (43.84)
  Double Blind Week 28- Tapering arm: number analyzed (Participants) | 16 | 61
  Double Blind Week 28- Tapering arm | -10.1 (24.28) | -3.8 (17.82)
  Double Blind Week 28- Withdrawal Arm: number analyzed (Participants) | 4 | 11
  Double Blind Week 28- Withdrawal Arm | -5.6 (45.59) | -17.2 (30.48)
  Double Blind Week 40- Tapering Arm: number analyzed (Participants) | 11 | 61
  Double Blind Week 40- Tapering Arm | -15.2 (33.53) | -4.4 (27.82)
  Double Blind Week 40- Withdrawal Arm: number analyzed (Participants) | 2 | 11
  Double Blind Week 40- Withdrawal Arm | -19.4 (27.50) | -16.2 (45.10)
  Flare Week 0- Tapering Arm: number analyzed (Participants) | 28 | 0
  Flare Week 0- Tapering Arm | -10.9 (39.82) |
  Flare Week 0- Withdrawal Arm: number analyzed (Participants) | 7 | 0
  Flare Week 0- Withdrawal Arm | -9.5 (38.05) |
  Flare Week 4- Tapering Arm: number analyzed (Participants) | 25 | 0
  Flare Week 4- Tapering Arm | -17.3 (40.07) |
  Flare Week 4- Withdrawal Arm: number analyzed (Participants) | 6 | 0
  Flare Week 4- Withdrawal Arm | -6.5 (48.23) |
  Flare Week 10- Tapering Arm: number analyzed (Participants) | 27 | 0
  Flare Week 10- Tapering Arm | -10.7 (44.07) |
  Flare Week 10- Withdrawal Arm: number analyzed (Participants) | 7 | 0
  Flare Week 10- Withdrawal Arm | 7.9 (34.23) |
  Flare Week 16- Tapering Arm: number analyzed (Participants) | 28 | 0
  Flare Week 16- Tapering Arm | -7.5 (25.49) |
  Flare Week 16- Withdrawal Arm: number analyzed (Participants) | 7 | 0
  Flare Week 16- Withdrawal Arm | -16.7 (39.67) |

32. Secondary Outcome: Mean Change From Double-blind Baseline in Treatment Satisfaction Questionnaire for Medication (TSQM) Side Effects Score
Description: as for outcome 31
Time Frame: At Weeks 4, 16, 28, and 40 and from Flare Week 0 to Flare Week 16
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Flared Participants | Non-Flared Participants
Number analyzed (Participants) | 46 | 74
units on a scale
  Double Blind Week 16- Tapering Arm: number analyzed (Participants) | 35 | 61
  Double Blind Week 16- Tapering Arm | -8.0 (17.25) | -0.5 (11.26)
  Double Blind Week 16- Withdrawal Arm: number analyzed (Participants) | 8 | 11
  Double Blind Week 16- Withdrawal Arm | 9.4 (20.04) | 2.8 (9.42)
  Double Blind Week 28- Tapering arm: number analyzed (Participants) | 16 | 61
  Double Blind Week 28- Tapering arm | -2.7 (12.28) | 1.1 (7.44)
  Double Blind Week 28- Withdrawal Arm: number analyzed (Participants) | 4 | 11
  Double Blind Week 28- Withdrawal Arm | 14.1 (28.13) | 2.8 (9.42)
  Double Blind Week 40- Tapering Arm: number analyzed (Participants) | 11 | 61
  Double Blind Week 40- Tapering Arm | -2.3 (14.86) | 1.1 (11.61)
  Double Blind Week 40- Withdrawal Arm: number analyzed (Participants) | 2 | 11
  Double Blind Week 40- Withdrawal Arm | 28.1 (39.77) | 2.8 (9.42)
  Flare Week 0- Tapering Arm: number analyzed (Participants) | 28 | 0
  Flare Week 0- Tapering Arm | -5.1 (15.96) |
  Flare Week 0- Withdrawal Arm: number analyzed (Participants) | 7 | 0
  Flare Week 0- Withdrawal Arm | 2.7 (7.09) |
  Flare Week 4- Tapering Arm: number analyzed (Participants) | 25 | 0
  Flare Week 4- Tapering Arm | -5.0 (19.52) |
  Flare Week 4- Withdrawal Arm: number analyzed (Participants) | 6 | 0
  Flare Week 4- Withdrawal Arm | 3.1 (7.65) |
  Flare Week 10- Tapering Arm: number analyzed (Participants) | 27 | 0
  Flare Week 10- Tapering Arm | -3.7 (13.90) |
  Flare Week 10- Withdrawal Arm: number analyzed (Participants) | 7 | 0
  Flare Week 10- Withdrawal Arm | 2.7 (7.09) |
  Flare Week 16- Tapering Arm: number analyzed (Participants) | 28 | 0
  Flare Week 16- Tapering Arm | -2.0 (6.60) |
  Flare Week 16- Withdrawal Arm: number analyzed (Participants) | 7 | 0
  Flare Week 16- Withdrawal Arm | 2.7 (7.09) |

33. Secondary Outcome: Mean Change From Double-blind Baseline in Treatment Satisfaction Questionnaire for Medication (TSQM) Convenience Score
Description: as for outcome 31
Time Frame: At Weeks 4, 16, 28, and 40 and from Flare Week 0 to Flare Week 16
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Flared Participants | Non-Flared Participants
Number analyzed (Participants) | 46 | 74
units on a scale
  Double Blind Week 16- Tapering Arm: number analyzed (Participants) | 35 | 61
  Double Blind Week 16- Tapering Arm | -0.2 (16.96) | 0.8 (13.45)
  Double Blind Week 16- Withdrawal Arm: number analyzed (Participants) | 8 | 11
  Double Blind Week 16- Withdrawal Arm | -4.9 (19.57) | 4.0 (10.86)
  Double Blind Week 28- Tapering arm: number analyzed (Participants) | 16 | 61
  Double Blind Week 28- Tapering arm | 0.0 (18.70) | -1.0 (15.47)
  Double Blind Week 28- Withdrawal Arm: number analyzed (Participants) | 4 | 11
  Double Blind Week 28- Withdrawal Arm | -4.2 (12.32) | -3.5 (13.21)
  Double Blind Week 40- Tapering Arm: number analyzed (Participants) | 11 | 61
  Double Blind Week 40- Tapering Arm | -4.0 (9.65) | -0.1 (16.50)
  Double Blind Week 40- Withdrawal Arm: number analyzed (Participants) | 2 | 11
  Double Blind Week 40- Withdrawal Arm | -16.7 (23.57) | 2.5 (18.32)
  Flare Week 0- Tapering Arm: number analyzed (Participants) | 28 | 0
  Flare Week 0- Tapering Arm | 4.2 (12.53) |
  Flare Week 0- Withdrawal Arm: number analyzed (Participants) | 7 | 0
  Flare Week 0- Withdrawal Arm | -7.1 (14.60) |
  Flare Week 4- Tapering Arm: number analyzed (Participants) | 25 | 0
  Flare Week 4- Tapering Arm | 4.4 (19.84) |
  Flare Week 4- Withdrawal Arm: number analyzed (Participants) | 6 | 0
  Flare Week 4- Withdrawal Arm | 5.6 (18.92) |
  Flare Week 10- Tapering Arm: number analyzed (Participants) | 27 | 0
  Flare Week 10- Tapering Arm | 1.2 (10.60) |
  Flare Week 10- Withdrawal Arm: number analyzed (Participants) | 7 | 0
  Flare Week 10- Withdrawal Arm | 0.8 (16.49) |
  Flare Week 16- Tapering Arm: number analyzed (Participants) | 28 | 0
  Flare Week 16- Tapering Arm | 1.6 (19.65) |
  Flare Week 16- Withdrawal Arm: number analyzed (Participants) | 7 | 0
  Flare Week 16- Withdrawal Arm | 0.8 (20.89) |

34. Secondary Outcome: Mean Change From Double-blind Baseline in Treatment Satisfaction Questionnaire for Medication (TSQM) Global Satisfaction Score
Description: as for outcome 31
Time Frame: At Weeks 4, 16, 28, and 40 and from Flare Week 0 to Flare Week 16
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Flared Participants | Non-Flared Participants
Number analyzed (Participants) | 46 | 74
units on a scale
  Double Blind Week 16- Tapering Arm: number analyzed (Participants) | 35 | 61
  Double Blind Week 16- Tapering Arm | -11.6 (24.99) | -3.4 (17.91)
  Double Blind Week 16- Withdrawal Arm: number analyzed (Participants) | 8 | 11
  Double Blind Week 16- Withdrawal Arm | -2.7 (15.24) | 0.6 (22.69)
  Double Blind Week 28- Tapering arm: number analyzed (Participants) | 16 | 61
  Double Blind Week 28- Tapering arm | -2.2 (12.70) | -5.7 (14.97)
  Double Blind Week 28- Withdrawal Arm: number analyzed (Participants) | 4 | 11
  Double Blind Week 28- Withdrawal Arm | 5.4 (15.84) | -4.5 (25.81)
  Double Blind Week 40- Tapering Arm: number analyzed (Participants) | 11 | 61
  Double Blind Week 40- Tapering Arm | -3.2 (13.31) | -2.6 (15.10)
  Double Blind Week 40- Withdrawal Arm: number analyzed (Participants) | 2 | 11
  Double Blind Week 40- Withdrawal Arm | 0.0 (10.10) | -3.2 (21.98)
  Flare Week 0- Tapering Arm: number analyzed (Participants) | 28 | 0
  Flare Week 0- Tapering Arm | -11.7 (27.58) |
  Flare Week 0- Withdrawal Arm: number analyzed (Participants) | 7 | 0
  Flare Week 0- Withdrawal Arm | -9.2 (25.66) |
  Flare Week 4- Tapering Arm: number analyzed (Participants) | 25 | 0
  Flare Week 4- Tapering Arm | -3.1 (20.32) |
  Flare Week 4- Withdrawal Arm: number analyzed (Participants) | 6 | 0
  Flare Week 4- Withdrawal Arm | -1.2 (24.08) |
  Flare Week 10- Tapering Arm: number analyzed (Participants) | 27 | 0
  Flare Week 10- Tapering Arm | -0.8 (13.77) |
  Flare Week 10- Withdrawal Arm: number analyzed (Participants) | 7 | 0
  Flare Week 10- Withdrawal Arm | -2.0 (18.77) |
  Flare Week 16- Tapering Arm: number analyzed (Participants) | 28 | 0
  Flare Week 16- Tapering Arm | -6.6 (24.20) |
  Flare Week 16- Withdrawal Arm: number analyzed (Participants) | 7 | 0
  Flare Week 16- Withdrawal Arm | -8.2 (16.72) |

35. Secondary Outcome: Mean Change From Double-blind Baseline in Work Productivity and Activity Impairment (WPAI) Overall Work Impairment and Activity Impairment Scores
Description: The Work Productivity and Activity Impairment (WPAI) questionnaire for general health is a validated tool in rheumatoid arthritis consisting of 6 questions, based on participant recall of the previous 7 days. WPAI assesses work time missed due to illness (absenteeism), impairment at work due to health (presenteeism), overall work impairment due to health (an aggregate measure of both absenteeism and presenteeism), and total non-occupational activity impairment due to health. WPAI scores are expressed as impairment percentages, with higher scores indicating worse outcomes. A negative change from baseline indicates improvement.
Time Frame: At Weeks 4, 28, and 40 and Flare Weeks 0, 10, and 16
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: percent impairment
Arm/Group | Flared Participants | Non-Flared Participants
Number analyzed (Participants) | 46 | 75
percent impairment
  Overall Work Impairment at Week 28- Tapering Arm: number analyzed (Participants) | 2 | 27
  Overall Work Impairment at Week 28- Tapering Arm | 15.0 (21.21) | 3.5 (10.68)
  Overall Work Impairment at Week 28- Withdrawal Arm: number analyzed (Participants) | 1 | 5
  Overall Work Impairment at Week 28- Withdrawal Arm | 0.0 | 0.6 (8.12)
  Activity Impairment at Week 28- Tapering arm: number analyzed (Participants) | 14 | 61
  Activity Impairment at Week 28- Tapering arm | 5.0 (19.51) | 2.8 (13.43)
  Activity Impairment at Week 28- Withdrawal Arm: number analyzed (Participants) | 3 | 11
  Activity Impairment at Week 28- Withdrawal Arm | 10.0 (17.32) | -0.9 (7.01)
  Overall Work Impairment at Week 40- Tapering Arm: number analyzed (Participants) | 0 | 28
  Overall Work Impairment at Week 40- Tapering Arm |  | 3.4 (18.78)
  Overall Work Impairment at Week 40- Withdrawal Arm: number analyzed (Participants) | 0 | 5
  Overall Work Impairment at Week 40- Withdrawal Arm |  | 0.6 (8.12)
  Activity Impairment at Week 40- Tapering arm: number analyzed (Participants) | 7 | 61
  Activity Impairment at Week 40- Tapering arm | 15.7 (9.76) | 0.5 (13.59)
  Activity Impairment at Week 40- Withdrawal Arm: number analyzed (Participants) | 1 | 11
  Activity Impairment at Week 40- Withdrawal Arm | 20.0 | 0.0 (6.32)
  Overall Work Impairment Flare Wk 0- Tapering Arm: number analyzed (Participants) | 5 | 0
  Overall Work Impairment Flare Wk 0- Tapering Arm | 14.0 (27.02) |
  Overall Work Impairment Flare Wk 0- Withdrawal Arm: number analyzed (Participants) | 2 | 0
  Overall Work Impairment Flare Wk 0- Withdrawal Arm | 5.0 (7.07) |
  Activity Impairment Flare Week 0- Tapering Arm: number analyzed (Participants) | 22 | 0
  Activity Impairment Flare Week 0- Tapering Arm | 25.9 (31.57) |
  Activity Impairment Flare Week 0- Withdrawal Arm: number analyzed (Participants) | 5 | 0
  Activity Impairment Flare Week 0- Withdrawal Arm | 8.0 (25.88) |
  Overall Work Impairment Flare Wk 10- Tapering Arm: number analyzed (Participants) | 8 | 0
  Overall Work Impairment Flare Wk 10- Tapering Arm | -0.2 (8.78) |
  Overall Work Impairment Flare W 10- Withdrawal Arm: number analyzed (Participants) | 2 | 0
  Overall Work Impairment Flare W 10- Withdrawal Arm | 5.0 (7.07) |
  Activity Impairment Flare Wk 10- Tapering Arm: number analyzed (Participants) | 26 | 0
  Activity Impairment Flare Wk 10- Tapering Arm | 6.5 (15.48) |
  Activity Impairment Flare W 10- Withdrawal Arm: number analyzed (Participants) | 7 | 0
  Activity Impairment Flare W 10- Withdrawal Arm | 12.9 (13.80) |
  Overall Work Impairment Flare Wk 16- Tapering Arm: number analyzed (Participants) | 8 | 0
  Overall Work Impairment Flare Wk 16- Tapering Arm | 10.0 (14.82) |
  Overall Work Impairment Flare W 16- Withdrawal Arm: number analyzed (Participants) | 3 | 0
  Overall Work Impairment Flare W 16- Withdrawal Arm | 10.0 (10.00) |
  Activity Impairment Flare Wk 16- Tapering Arm: number analyzed (Participants) | 29 | 0
  Activity Impairment Flare Wk 16- Tapering Arm | 11.0 (17.39) |
  Activity Impairment Flare Wk 16- Withdrawal Arm: number analyzed (Participants) | 8 | 0
  Activity Impairment Flare Wk 16- Withdrawal Arm | 8.8 (11.26) |

36. Secondary Outcome: Mean Change From Double-blind Baseline in Short-Form 36 Version 2 Health Survey (SF-36v2) Physical Component Summary (PCS) Score
Description: The SF-36v2 is a non-disease specific Health Related Quality of Life (HRQoL) instrument. The SF-36v2 comprises 36 total items (questions) targeting a subject's functional health and well-being in 8 domains (physical functioning, role physical, bodily pain, general health, vitality, social functioning, role emotional and mental health) with a recall period of four weeks. Domain scores are aggregated into a Physical Component Summary (PCS) score and a Mental Component Summary (MCS) score. SF-36v2 scores for each domain and PCS/MCS range from 0-100: higher scores indicate a better state of health and a decrease from baseline represents worsening.
Time Frame: At Weeks 4, 28, and 40 and from Flare Week 0 to Flare Week 16
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Flared Participants | Non-Flared Participants
Number analyzed (Participants) | 45 | 74
units on a scale
  Double Blind Week 28- Tapering arm: number analyzed (Participants) | 13 | 60
  Double Blind Week 28- Tapering arm | -2.9 (7.53) | -1.1 (4.18)
  Double Blind Week 28- Withdrawal Arm: number analyzed (Participants) | 3 | 11
  Double Blind Week 28- Withdrawal Arm | -1.9 (7.39) | -2.4 (3.97)
  Double Blind Week 40- Tapering Arm: number analyzed (Participants) | 6 | 60
  Double Blind Week 40- Tapering Arm | -5.5 (6.42) | -0.4 (5.53)
  Double Blind Week 40- Withdrawal Arm: number analyzed (Participants) | 1 | 11
  Double Blind Week 40- Withdrawal Arm | -1.6 | -2.1 (5.22)
  Flare Week 0- Tapering Arm: number analyzed (Participants) | 22 | 0
  Flare Week 0- Tapering Arm | -10.8 (10.85) |
  Flare Week 0- Withdrawal Arm: number analyzed (Participants) | 5 | 0
  Flare Week 0- Withdrawal Arm | -2.4 (10.81) |
  Flare Week 4- Tapering Arm: number analyzed (Participants) | 24 | 0
  Flare Week 4- Tapering Arm | -5.2 (8.37) |
  Flare Week 4- Withdrawal Arm: number analyzed (Participants) | 6 | 0
  Flare Week 4- Withdrawal Arm | -8.0 (7.35) |
  Flare Week 10- Tapering Arm: number analyzed (Participants) | 25 | 0
  Flare Week 10- Tapering Arm | -4.0 (7.22) |
  Flare Week 10- Withdrawal Arm: number analyzed (Participants) | 7 | 0
  Flare Week 10- Withdrawal Arm | -4.0 (4.57) |
  Flare Week 16- Tapering Arm: number analyzed (Participants) | 28 | 0
  Flare Week 16- Tapering Arm | -3.8 (7.38) |
  Flare Week 16- Withdrawal Arm: number analyzed (Participants) | 7 | 0
  Flare Week 16- Withdrawal Arm | -2.5 (2.80) |

37. Secondary Outcome: Mean Change From Double-blind Baseline in Short-Form 36 Version 2 Health Survey (SF-36v2) Mental Component Summary (MCS) Score
Description: as for outcome 36
Time Frame: At Weeks 4, 28, and 40 and from Flare Week 0 to Flare Week 16
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Flared Participants | Non-Flared Participants
Number analyzed (Participants) | 45 | 74
units on a scale
  Double Blind Week 28- Tapering arm: number analyzed (Participants) | 13 | 60
  Double Blind Week 28- Tapering arm | -5.5 (11.31) | -0.8 (6.02)
  Double Blind Week 28- Withdrawal Arm: number analyzed (Participants) | 3 | 11
  Double Blind Week 28- Withdrawal Arm | -5.2 (5.90) | -0.1 (7.20)
  Double Blind Week 40- Tapering Arm: number analyzed (Participants) | 6 | 60
  Double Blind Week 40- Tapering Arm | -3.5 (11.14) | -0.8 (5.89)
  Double Blind Week 40- Withdrawal Arm: number analyzed (Participants) | 1 | 11
  Double Blind Week 40- Withdrawal Arm | -8.5 | -0.4 (6.71)
  Flare Week 0- Tapering Arm: number analyzed (Participants) | 22 | 0
  Flare Week 0- Tapering Arm | -4.1 (11.43) |
  Flare Week 0- Withdrawal Arm: number analyzed (Participants) | 5 | 0
  Flare Week 0- Withdrawal Arm | 0.4 (4.59) |
  Flare Week 4- Tapering Arm: number analyzed (Participants) | 24 | 0
  Flare Week 4- Tapering Arm | -2.0 (5.95) |
  Flare Week 4- Withdrawal Arm: number analyzed (Participants) | 6 | 0
  Flare Week 4- Withdrawal Arm | -0.5 (2.51) |
  Flare Week 10- Tapering Arm: number analyzed (Participants) | 25 | 0
  Flare Week 10- Tapering Arm | -1.1 (10.14) |
  Flare Week 10- Withdrawal Arm: number analyzed (Participants) | 7 | 0
  Flare Week 10- Withdrawal Arm | -0.4 (3.06) |
  Flare Week 16- Tapering Arm: number analyzed (Participants) | 28 | 0
  Flare Week 16- Tapering Arm | -4.0 (11.01) |
  Flare Week 16- Withdrawal Arm: number analyzed (Participants) | 7 | 0
  Flare Week 16- Withdrawal Arm | 0.1 (2.55) |

38. Secondary Outcome: Mean Change From Double-blind Baseline in Functional Assessment of Chronic Illness Therapy (FACIT) Fatigue Scale
Description: The FACIT-Fatigue questionnaire is a participant questionnaire that consists of 13 questions designed to measure the degree of fatigue experienced by participants in the previous 7 days. Participants respond to the questions on a scale from 'not at all' (0) to 'very much' (4). The scale score is computed by summing the item scores, after reversing those items that are worded in the negative direction. The FACIT-Fatigue subscale score ranges from 0 to 52, where higher scores represent less fatigue. A negative change from baseline indicates worsening.
Time Frame: At Weeks 4, 16, 28, and 40 and from Flare Week 0 to Flare Week 16
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Flared Participants | Non-Flared Participants
Number analyzed (Participants) | 46 | 74
units on a scale
  Double Blind Week 16- Tapering Arm: number analyzed (Participants) | 35 | 61
  Double Blind Week 16- Tapering Arm | -6.0 (9.80) | -1.5 (5.42)
  Double Blind Week 16- Withdrawal Arm: number analyzed (Participants) | 9 | 11
  Double Blind Week 16- Withdrawal Arm | -2.3 (3.39) | -1.9 (3.27)
  Double Blind Week 28- Tapering arm: number analyzed (Participants) | 16 | 61
  Double Blind Week 28- Tapering arm | -3.5 (7.58) | -1.6 (5.60)
  Double Blind Week 28- Withdrawal Arm: number analyzed (Participants) | 4 | 11
  Double Blind Week 28- Withdrawal Arm | -4.3 (7.23) | -2.2 (4.67)
  Double Blind Week 40- Tapering Arm: number analyzed (Participants) | 11 | 61
  Double Blind Week 40- Tapering Arm | -6.4 (8.44) | -0.4 (4.00)
  Double Blind Week 40- Withdrawal Arm: number analyzed (Participants) | 2 | 11
  Double Blind Week 40- Withdrawal Arm | -2.5 (6.36) | -1.5 (4.78)
  Flare Week 0- Tapering Arm: number analyzed (Participants) | 28 | 0
  Flare Week 0- Tapering Arm | -7.4 (11.17) |
  Flare Week 0- Withdrawal Arm: number analyzed (Participants) | 8 | 0
  Flare Week 0- Withdrawal Arm | -3.6 (4.75) |
  Flare Week 4- Tapering Arm: number analyzed (Participants) | 25 | 0
  Flare Week 4- Tapering Arm | -3.8 (9.19) |
  Flare Week 4- Withdrawal Arm: number analyzed (Participants) | 6 | 0
  Flare Week 4- Withdrawal Arm | -4.7 (5.43) |
  Flare Week 10- Tapering Arm: number analyzed (Participants) | 27 | 0
  Flare Week 10- Tapering Arm | -3.9 (8.44) |
  Flare Week 10- Withdrawal Arm: number analyzed (Participants) | 7 | 0
  Flare Week 10- Withdrawal Arm | -2.4 (4.47) |
  Flare Week 16- Tapering Arm: number analyzed (Participants) | 28 | 0
  Flare Week 16- Tapering Arm | -4.5 (9.01) |
  Flare Week 16- Withdrawal Arm: number analyzed (Participants) | 7 | 0
  Flare Week 16- Withdrawal Arm | -1.7 (1.89) |

39. Secondary Outcome: Mean Change From Double-blind Baseline in Serum Levels of C-reactive Protein (CRP)
Description: C-Reactive Protein (CRP; mg/L) was measured from blood samples as a marker for inflammation. Higher levels are indicative of more inflammation. Negative values indicate improvement from baseline.
Time Frame: From Week 4 to Week 40 and from Flare Week 0 to Flare Week 16
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mg/L
Arm/Group | Flared Participants | Non-Flared Participants
Number analyzed (Participants) | 46 | 76
mg/L
  Double Blind Week 10- Tapering Arm: number analyzed (Participants) | 36 | 64
  Double Blind Week 10- Tapering Arm | -7.9 (48.87) | 1.7 (12.92)
  Double Blind Week 10- Withdrawal Arm: number analyzed (Participants) | 9 | 11
  Double Blind Week 10- Withdrawal Arm | -0.2 (3.55) | -0.6 (2.53)
  Double Blind Week 16- Tapering Arm: number analyzed (Participants) | 35 | 63
  Double Blind Week 16- Tapering Arm | -7.4 (49.77) | -0.4 (4.26)
  Double Blind Week 16- Withdrawal Arm: number analyzed (Participants) | 9 | 11
  Double Blind Week 16- Withdrawal Arm | 6.6 (12.26) | -0.1 (3.67)
  Double Blind Week 22- Tapering Arm: number analyzed (Participants) | 19 | 63
  Double Blind Week 22- Tapering Arm | 3.6 (9.69) | -0.0 (5.43)
  Double Blind Week 22- Withdrawal arm: number analyzed (Participants) | 4 | 11
  Double Blind Week 22- Withdrawal arm | 0.6 (0.37) | -0.9 (3.38)
  Double Blind Week 28- Tapering arm: number analyzed (Participants) | 16 | 63
  Double Blind Week 28- Tapering arm | 0.5 (3.85) | -0.4 (4.65)
  Double Blind Week 28- Withdrawal Arm: number analyzed (Participants) | 4 | 11
  Double Blind Week 28- Withdrawal Arm | 1.1 (1.34) | 2.5 (11.60)
  Double Blind Week 34- Tapering Arm: number analyzed (Participants) | 12 | 63
  Double Blind Week 34- Tapering Arm | 3.2 (10.13) | -0.4 (4.41)
  Double Blind Week 34- Withdrawal Arm: number analyzed (Participants) | 2 | 11
  Double Blind Week 34- Withdrawal Arm | 1.8 (1.89) | 0.3 (5.98)
  Double Blind Week 40- Tapering Arm: number analyzed (Participants) | 11 | 63
  Double Blind Week 40- Tapering Arm | 1.0 (5.69) | -0.3 (4.18)
  Double Blind Week 40- Withdrawal Arm: number analyzed (Participants) | 2 | 11
  Double Blind Week 40- Withdrawal Arm | 8.3 (11.60) | -0.1 (3.43)
  Flare Week 0- Tapering Arm: number analyzed (Participants) | 30 | 0
  Flare Week 0- Tapering Arm | -7.4 (54.12) |
  Flare Week 0- Withdrawal Arm: number analyzed (Participants) | 8 | 0
  Flare Week 0- Withdrawal Arm | 5.4 (12.67) |
  Flare Week 4- Tapering Arm: number analyzed (Participants) | 30 | 0
  Flare Week 4- Tapering Arm | -8.5 (55.47) |
  Flare Week 4- Withdrawal Arm: number analyzed (Participants) | 8 | 0
  Flare Week 4- Withdrawal Arm | -1.3 (4.01) |
  Flare Week 10- Tapering Arm: number analyzed (Participants) | 30 | 0
  Flare Week 10- Tapering Arm | -9.5 (55.61) |
  Flare Week 10- Withdrawal Arm: number analyzed (Participants) | 8 | 0
  Flare Week 10- Withdrawal Arm | -0.6 (0.97) |
  Flare Week 16- Tapering Arm: number analyzed (Participants) | 30 | 0
  Flare Week 16- Tapering Arm | -9.1 (53.70) |
  Flare Week 16- Withdrawal Arm: number analyzed (Participants) | 8 | 0
  Flare Week 16- Withdrawal Arm | -0.8 (2.74) |

40. Secondary Outcome: Mean Change From Double-blind Baseline in Serum Levels of Erythrocyte Sedimentation Rate (ESR)
Description: Erythrocyte sedimentation rate (ESR; mm/hour) indirectly measures how much inflammation is in the body. A higher ESR is indicative of increased inflammation. Negative values indicate improvement from baseline.
Time Frame: From Week 4 to Week 40 and from Flare Week 0 to Flare Week 16
Population: as for outcome 10
Measure: Mean (Standard Deviation); unit: mm/hour
Arm/Group | Flared Participants | Non-Flared Participants
Number analyzed (Participants) | 46 | 76
mm/hour
  Double Blind Week 10- Tapering Arm: number analyzed (Participants) | 37 | 64
  Double Blind Week 10- Tapering Arm | 4.1 (11.25) | 0.7 (5.22)
  Double Blind Week 10- Withdrawal Arm: number analyzed (Participants) | 9 | 11
  Double Blind Week 10- Withdrawal Arm | 0.9 (9.24) | -1.5 (5.43)
  Double Blind Week 16- Tapering Arm: number analyzed (Participants) | 35 | 63
  Double Blind Week 16- Tapering Arm | 4.6 (10.73) | 0.5 (5.82)
  Double Blind Week 16- Withdrawal Arm: number analyzed (Participants) | 9 | 11
  Double Blind Week 16- Withdrawal Arm | 5.2 (15.23) | -0.3 (5.31)
  Double Blind Week 22- Tapering Arm: number analyzed (Participants) | 19 | 63
  Double Blind Week 22- Tapering Arm | 3.5 (10.73) | -0.5 (7.38)
  Double Blind Week 22- Withdrawal arm: number analyzed (Participants) | 4 | 11
  Double Blind Week 22- Withdrawal arm | 2.8 (9.22) | -0.3 (4.22)
  Double Blind Week 28- Tapering arm: number analyzed (Participants) | 16 | 63
  Double Blind Week 28- Tapering arm | 3.4 (8.18) | 0.4 (6.93)
  Double Blind Week 28- Withdrawal Arm: number analyzed (Participants) | 4 | 11
  Double Blind Week 28- Withdrawal Arm | 6.0 (10.10) | 1.0 (5.04)
  Double Blind Week 34- Tapering Arm: number analyzed (Participants) | 12 | 63
  Double Blind Week 34- Tapering Arm | 4.8 (7.28) | 0.3 (7.57)
  Double Blind Week 34- Withdrawal Arm: number analyzed (Participants) | 2 | 11
  Double Blind Week 34- Withdrawal Arm | -5.0 (1.41) | -0.5 (5.94)
  Double Blind Week 40- Tapering Arm: number analyzed (Participants) | 11 | 63
  Double Blind Week 40- Tapering Arm | 10.2 (13.22) | 1.4 (7.19)
  Double Blind Week 40- Withdrawal Arm: number analyzed (Participants) | 2 | 11
  Double Blind Week 40- Withdrawal Arm | -2.0 (5.66) | 4.7 (8.89)
  Flare Week 0- Tapering Arm: number analyzed (Participants) | 30 | 0
  Flare Week 0- Tapering Arm | 10.4 (12.50) |
  Flare Week 0- Withdrawal Arm: number analyzed (Participants) | 8 | 0
  Flare Week 0- Withdrawal Arm | 13.0 (11.90) |
  Flare Week 4- Tapering Arm: number analyzed (Participants) | 30 | 0
  Flare Week 4- Tapering Arm | 7.2 (9.82) |
  Flare Week 4- Withdrawal Arm: number analyzed (Participants) | 8 | 0
  Flare Week 4- Withdrawal Arm | 8.5 (9.52) |
  Flare Week 10- Tapering Arm: number analyzed (Participants) | 30 | 0
  Flare Week 10- Tapering Arm | 5.8 (10.16) |
  Flare Week 10- Withdrawal Arm: number analyzed (Participants) | 8 | 0
  Flare Week 10- Withdrawal Arm | 4.4 (6.91) |
  Flare Week 16- Tapering Arm: number analyzed (Participants) | 30 | 0
  Flare Week 16- Tapering Arm | 8.0 (10.95) |
  Flare Week 16- Withdrawal Arm: number analyzed (Participants) | 8 | 0
  Flare Week 16- Withdrawal Arm | 7.0 (14.40) |

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) and serious adverse events (TESAEs) were collected from first dose of study drug until 70 days after the last dose of study drug in the Double-blind Period (up to 50 weeks); for participants who experienced flare during the double-blind period, AEs were collected until 70 days after the last dose of study drug in the 16-week Open-label Rescue Period (up to 66 weeks).
Description: TEAEs and TESAEs are defined as any adverse event (AE) with an onset date that is on or after the first dose of study drug until 70 days after the last dose of study drug and were collected whether elicited or spontaneously reported by the participant.
Groups:
- Adalimumab 40 mg Eow: 40 mg adalimumab administered subcutaneously every other week (eow) from Week 0 to Week 4
Arm/Group | Adalimumab 40 mg Eow | Adalimumab Tapering | Adalimumab Withdrawal Arm | Adalimumab 40 mg Eow Rescue Arm
All-Cause Mortality (participants affected / at risk) | 0/146 | 0/102 | 0/20 | 0/39
Serious Adverse Events (participants affected / at risk) | 4/146 | 1/102 | 0/20 | 3/39
Other Adverse Events (participants affected / at risk) | 11/146 | 33/102 | 12/20 | 13/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adalimumab 40 mg Eow (N=146) | Adalimumab Tapering (N=102) | Adalimumab Withdrawal Arm (N=20) | Adalimumab 40 mg Eow Rescue Arm (N=39)
ATRIAL FIBRILLATION (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
RETINAL VEIN OCCLUSION (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COMMINUTED FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TRANSIENT ISCHAEMIC ATTACK (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Adalimumab 40 mg Eow (N=146) | Adalimumab Tapering (N=102) | Adalimumab Withdrawal Arm (N=20) | Adalimumab 40 mg Eow Rescue Arm (N=39)
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
INFLUENZA (Infections and infestations) | 0 (0) | 5 (6) | 2 (2) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 3 (3) | 1 (1) | 1 (1)
NASOPHARYNGITIS (Infections and infestations) | 4 (4) | 16 (17) | 4 (5) | 4 (4)
PHARYNGOTONSILLITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TONSILLITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
TOOTH INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
URINARY TRACT INFECTION (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
LIMB INJURY (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
C-REACTIVE PROTEIN INCREASED (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
HEPATIC ENZYME INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 6 (10) | 0 (0) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OSTEOPOROSIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 5 (5) | 1 (1) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4 (4) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2016-02-25): https://cdn.clinicaltrials.gov/large-docs/51/NCT02198651/Prot_000.pdf
  • Statistical Analysis Plan (2018-07-19): https://cdn.clinicaltrials.gov/large-docs/51/NCT02198651/SAP_001.pdf